# **Study Protocol**

Study Title: Akashic Records and Mental Health Outcomes

ClinicalTrials.gov Identifier: NCTXXXXXXX

Document Type: Study Protocol

Revision Date: [5.21.24]

Principal Investigator: Candice S. Rasa, LCSW

Co-Investigator: Sarah Coleman, LCSW

Sponsor: Rasa Healing, Inc.

#### **STUDY TITLE:**

Akashic Records and Mental Health Outcomes

#### PRINCIPAL INVESTIGATOR:

Name: Candice S. Rasa, LCSW, Sponsor

#### **CO-INVESTIGATORS:**

Name: Sarah Coleman, LCSW, Independent Evaluator

# **SPONSOR:**

Rasa Healing Services, Inc.

## **VERSION/DATE:**

Version 3 05/21/24

Check any **applicable** boxes in the table below – you will be asked for further detail on these topics later in the protocol:

| Indicate Vulnerable Population(s) to be Enrolled | ☐ Children ☐ Cognitively Impaired Adults ☐ Pregnant Women (IF the research activities will affect the pregnancy or the fetus) ☐ Prisoners (or other detained/paroled individuals) n/a |
|---|---|
| Research has U.S. Federal<br>government funding (e.g.,<br>NIH, NSF, other federal<br>agencies/departments) | □<br>n/a |

#### TABLE OF CONTENTS

- 1. Purpose of the study
- 2. Background/ literature review/ rationale for the study
- 3. Inclusion and Exclusion criteria
- 4. Sample size
- 5. Recruitment and Screening Methods
  - a. Recruitment Process
  - b. Prescreening and screening process
  - c. Prescreen and Enrollment Checklist
  - d. Prescreen Script
- 6. Research locations

- 7. Multi-site Research (research that involves external collaborating institutions and individuals)
- 8. Procedures Involved
  - a. Akashic Records Reader Methods
  - b. Akashic Channeling
  - c. Akashic Record Channeling Verses Therapy
  - d. Akashic Records Procedure
  - e. Estimated Time Commitment
  - f. Self-Report Assessments
  - g. Semi Structured Interview
  - h. Semi-Structured Interview Script and Questions
- 9. Research with Vulnerable Populations
- 10. Incomplete Disclosure or Deception
- 11. Consent Process
- 12. Research with Children Parental Permission, Child Assent, and Other Considerations
- 13. Waiver of Participant Signature on Consent Form
- 14. Waivers and Alterations of Consent Information
- 15. Financial Compensation
- 16. Audio/Video Recording/Photography:
- 17. Potential Benefits of this Research
- 18. Risk to Participants
- 19. Provisions to Protect Participant Privacy and Data Confidentiality
  - a. Participant Privacy
  - b. Confidentiality of Data and Biospecimens
- 20. Data Monitoring Plan to Ensure Safety of Participants
- 21. Long-term Data and Specimen Storage and Sharing
- 22. Qualifications of Research Team to Conduct Research
- 23. References

# **Appendix A- Procedures**

- i. Standard Operating Procedure for Participant Identification and Recruitment
- ii. Standard Operating Procedure for Participant Eligibility Confirmation
- iii. Standard Operating Procedure for Participant Enrollment
- iv. Standard Operating Procedure for Assigning Unique Identification Numbers
- v. Standard Operating Procedure for Recording and Storage of Akashic Sessions
- vi. Standard Operating Procedure for Participant Completion of Clinical Scales
- vii. Standard Operating Procedure for Scheduling, Recording, and Storing Virtual Interviews
- viii. Standard Operating Procedure for Qualitative Analysis of Structured Interviews
- ix. Standard Operating Procedure for Managing Conflict of Interest in a Study Measuring the Effectiveness of Akashic Record Sessions
- x. Standard Operating Procedure for Participant Withdrawal from Study

## **Appendix B- Scripts**

- i. Prescreen scripts
- ii. Akashic scripts
- iii. Semi-structured scripts

# **Appendix C- Staff Checklists**

- i. Phase 1: Application and Approval Process
- ii. Phase 2: Self Assessments and Akashic Session
- iii. Phase 3: Final Assessments and Semi-structured Interview

# **Appendix D- Templates**

- i. Recruitment Templates
  - a. Landing Page + Email marketing
  - b. Social Media posts
- ii. Email Sequence Templates
- iii. Akashic Prep Template
- iii. Mental Health Referral Template

# 1. Purpose of the study:

The purpose of this study is to investigate whether Akashic Records sessions, facilitated by Candice Rasa, LCSW, contribute to improvements in mental health outcomes. More specifically, we are studying how 2 Akashic Record sessions impact mental health symptoms through self-report assessments. The self-report assessments include measuring levels of depression, anxiety and stress pre- and post-session. They also include measuring levels of resiliency and feelings of connectedness with oneself, their community, and all of humanity. The research question for this study is: Do Akashic Records sessions improve mental health outcomes as evidenced by a decrease in self-reported stress, anxiety and depression and/or an increase in resiliency and connectedness?

# 2. Background / Literature Review / Rationale for the study:

#### Introduction

Transpersonal theory has grown since the 1960's due to expansion of consciousness, the birth of humanistic psychology, Eastern philosophies and practices and pioneering figures. Transpersonal psychology involves the clinician assisting the client in achieving higher levels of being, from their current selves or trauma-flooded selves, to the "unitive self or real self" (Cowley, 1993, p.527). The Akashic Records are an energetic, nonphysical, cosmic, conscious, fluid, energy field that houses the ancestral and karmic information of all souls (Laszlo, 2021). Having your Akashic Records read can induce altered states of consciousness that may generate feelings of oneness, connection, love, and unity. Clients experiencing Akashic Records can have a transpersonal experience which may include a sudden clarity on life problems, objectivity, emotional integration, feelings of empowerment, and awareness of strengths, among other benefits. The shifts experienced during these sessions are believed to catalyze lasting

transformations, as Charles Tart suggests in his book *Altered states of consciousness*: "Research correlating mystical experience with improved psychological functioning does indeed suggest that people may undergo trait changes as a result of state changes." (Winter, 1999. P 18). Accessing the Akashic field in a therapeutic setting or measuring the impact of Akashic Records on client outcomes—specifically, mental health symptoms—has never been researched or examined before despite growing public and professional interest in transpersonal methods. While research exists in demonstrating the benefits of altered states of consciousness to client mental health improvement, there is a gap in understanding howAkashic Records might impact mental health symptoms.

# Transpersonal Theory Roots

Transpersonal theory is based on clients achieving happiness, connection, purpose, love, and unity outside, or independent, of human experiences. Carl Jung (Swiss psychologist and psychoanalyst), Abraham Maslow (American Psychologist), and Stanislav Grof (Czech psychiatrist) are well known thought leaders in the mental health field that have initiated research, formalized protocol, and published articles highlighting the value of transpersonal theory in therapy. Transpersonal interventions in therapy place greater focus on altered states of consciousness, from which a client can see themselves and their lives from a transcended state. Elements researched in meta-analyses that define transpersonal modalities include "(a) states of consciousness, (b) highest or ultimate potential, (c) beyond ego or personal self, (d) transcendence, and (e) spiritual." (Lajoie and Shapiro, 1992, p 90). In the 1970's, humanistic psychology surged, and psychedelics were among the primary tools of transpersonal therapists, but recently, breathwork, hypnotherapy, and transcendental meditation, among others, have been studied.

#### Benefits of Transpersonal Interventions

There are many benefits to transpersonal interventions in practice settings. Transpersonal tools can be highly useful for clients experiencing extreme life transition and loss often associated with the human experience. It can "promote respect for self-determination while empowering and facilitating bio-psycho-social-spiritual growth." (Canda and Smith, 2001, p 64). Viktor Frankel, respected psychiatrist, Holocaust survivor, international author of *Man's Search for Meaning* and creator of logotherapy suggests that human suffering is relative in relation to the person's capacity to discern meaning or identify "a larger why" within his/her suffering (Frankel, 1946). As reported in case study examples, those in Holocaust concentration camps that did not experience purpose, meaning, or hope in relation to their condition not only experienced worsening mental health symptoms, but also died of unknown causes sooner than those who subscribed to transpersonal theories (Frankel, 1946). The backbone of transpersonal work is the "recognition, understanding, and realization of intuitive, spiritual, and transcendent states of consciousness" (Lajoie and Shapiro, 1992, p 91). This consciousness provides a larger, zoomed-out perspective from one's current state of emotional suffering or hardship, and may enable clients to adapt with greater resiliency to their current conditions.

There also exists an ongoing trend in the mental health field to include client spirituality as a necessary component in therapy due to client preference, desire, and comfort. Over "two-thirds of Americans prefer to collaborate with a mental health professional who maintains

religious and spiritual beliefs and values when they are seeking services about serious problems" (Lehman, 1993). At the National Multicultural Conference and Summit hosted by the American Psychological Association, Plante (2008) stated, "spirituality is a necessary condition for a psychology of human existence". Not only are clients preferring to include transpersonal discussion as part of their therapeutic process, but there is evidence of improved physical and emotional wellbeing as a result. Specifically, "those engaged and active with spiritual matters tend to be healthier, happier, have better habits, and more social support than those who are not" (Plante, 2008). Due to growing momentum towards spirituality as a fundamental component of psychological well being, there is a need for more evidence-based research on interventions within the transpersonal framework.

#### Mental Health Outcomes and Transpersonal Research

There are studies that reflect the benefits of transpersonal intervention to client emotional health. In one study looking at the reduction of fear in cancer patients, it was found that counseling based on transpersonal interventions reduced the fear and stress of cancer recurrence statistically in comparison to a control group (Sajadian, Zahrakar & Asadpour, 2021). Moreover, transpersonal methods also increased client relaxation, reduction of stress, and contributed to overall quality of life (Sajadian, Zahrakar & Asadpour).

In another study with 24 undergraduate students who underwent past life imagery, those who received a suggestion to engage a past life memory had better scores on certain sections of the psychological wellbeing scale versus those who received an open suggestion during the imagery. Also, all students who experienced guided imagery also reported increased transpersonal beliefs as a result of participating in the study. This suggests the power of transcendent interventions with increased mental health benefits for those who engaged in past life memory recall (Woods and Baruss, 2004).

In a study looking at 133 adult men with a tendency towards violence revealed that treatment for aggressive behavior was more effective when it included transpersonal dialogue, archetypal recognition, and emphasis on existential and religious wellbeing. They also discovered that "regardless of their ethnic identity, men sought to experience spiritual development at three different levels of consciousness: ego, soul, and spirit" (Dexter and Freeman, 2001).

Research examining another transpersonal tool—holotropic breathwork—also demonstrates positive results for reducing anxiety symptoms. In a meta-analysis evaluating the efficacy of breathwork in lowering levels of self-reported/subjective stress compared to non-breathwork controls were promising. Over 12 randomized controlled studies which included a total of 785 adults reflected "small to medium effects of lower levels of stress than control conditions" (Fincham, et al. 2023).

#### What are the Akashic Records?

The Akashic Records is a nonphysical, etheric, fluid, cosmic energy field where all occurrences are stored. The Akasha can also be explained as a sacred library, God's remembering, or the book of life (Todeschi, 1998) that houses soul memories or experiences.

Akasha itself, is a Sanskrit word for "ether" or all pervasive space. Scientists Nikola Tesla, David Bohm, and Harold Puthoff surmised "interactions in the domains of nature as well as of mind are mediated by a fundamental information field at the heart of the universe" (Laszlo, 2004, p 46). On a micro level, the Akasha is explained through quantum physics and specifically, the quantum vacuum as a "zero-point field." Scientists have looked at how nature's information can be tracked in this field and that everything that takes place in it, can be referred to its origin. For example, around the nineteenth century, quantum concepts such as "nonlocality" and "entanglement" became widely accepted through validated research. Specifically, information from one particle is transferred to another particle permanently (entanglement) and that memory is kept across all physical and time space barriers (nonlocality). "Every particle that has ever occupied the same quantum state as another particle remains correlated with it in a mysterious, non-energetic way...and maintains such connection despite distance measurement in millimeters or light years or time measurement of seconds or millions of years" (Laszlo, 2004, p34, p45). Ervin Laszlo, philosopher of science, integral theorist, author of over a dozen publications and books on the Akashic field and quantum consciousness stated that the Akasha is "the enduring record of all that happens and has ever happened, in space and time" (Laszlo, 2004). Laszlo is the grandfather of the "connectivity hypothesis," the concept that everything remains permanently and holographically recorded on a subquantum level and that as such, can be read, observed and viewed

#### Akashic Records in Human Sciences

Since the 1930's, scientists theorized the conceptual Akasha through quantum research, but physicians and counselors also utilized this energy field for the transpersonal benefits of clients seeking physical and emotional healing. Specifically, the Akashic field is accessed to relay past lifetimes and ancestral memories to clients who are struggling to integrate traumas stemming from nonlocal time and space that create deeply rooted emotional and physical suffering. There are several thought leaders who have documented the value of the Akasha in its use as a transpersonal tool. In the 1830's, Helena Petrovna Blavatsky, mystic, author of *Alchemy* and the Secret Doctrine, and founder of the Theosophical Society states this about the Akashic field: "It is the quintessence of all possible forms of energy, material, psychic, or spiritual; and contains within itself the germs of universal creation, which sprout forth under the impulse of the Divine Spirit." (Todeschi, 1998, p xiv). She theorized the Akasha as a valuable search tool for soul understanding and spiritual actualization. By using the Akashic field to examine one's life, we can perceive our divine nature. Rudolf Steiner, philosopher, educator, author of Cosmic Memory, and founder of Anthroposophical Society states that it is possible for those to read and discern the "Akashic Chronicle." Specifically, "the one who acquires the ability to perceive in the spiritual world comes to know past events in their eternal character (past lifetimes). They do not stand before him like the dead testimony of history but appear in full life" (Todeschi, 1998, p xv). Steiner used his psychic skills to connect to the Akashic field and encouraged other healers in helping roles to do the same. "Man can penetrate to the eternal origins of the things which vanish with time...a man broadens his power of cognition... and sees events which are not perceptible to the senses" (Todeschi, 1998, p xiv).

However, the most well known mystic who documented use of the Akashic field in human sciences was the Christian physician and founder of the Association for Research and Enlightenment, Edgar Cayce. He documented 40 years of client case studies where he

specifically channeled the Akashic Record for clients as a tool to alleviate emotional and physical distress. Edgar Cayce documented the purpose of the Akasha as "keeping track of and assisting with each soul's personal growth and transformation" (Todeschi, 1998, p5). Cayce noted that people he served were seeking meaning, purpose, explanation of traumas, and reprieve from suffering. He surmised that "God is essentially love, and the Universe is completely orderly" (Todeschi, 1998, p 5) and that each person on the planet had a specific purpose to achieve through a collection of experiences. He wrote meticulous transcriptions of sessions including numerous past life channelings for clients. Cayce wrote about positive client outcomes as a result of using Akashic information in sessions with people including: relationship healing, releasing entangled ancestral dynamics, clarity in decision-making, understanding of circumstances, feedback on possible outcomes or healthy choices, awareness of karmic debts, and identification of cyclical patterns. (Todeschi, 1998). Laszlo, Grof, Weiss, Cayce, and others, have been drawing a connection from the Akashic field to C.G. Jung's collective unconscious by utilizing the Akashic field for the purpose of soul-level healing.

#### Akashic Field and Past Life Memories

Stanislov Grof, M.D. and psychiatrist, is one of the leading conceptualizers of transpersonal psychology research and its use of non-ordinary states of consciousness for purposes of psychological healing, deep self-exploration, and obtaining growth and insights into the human psyche. "The existence of past-life experiences with all their remarkable characteristics is an unquestionable fact that can be verified by any serious researcher who is sufficiently open-minded and interested to check the evidence" (Grov, p 18). Grov noted several consistent "anomalous phenomena" or occurrences of client detailed memory to events and behaviors outside of their race, culture, and time when in altered states that were later validated with historical data.

Grov has published several articles detailing case studies of past life and karmic explorations with therapy clients. Grov discerned that individuals can access their past lifetimes in such altered states via the Akashic field. "The observations from the research of holotropic states suggest that the individual human psyche has – at least potentially – the capacity of accessing all the information stored in the Akashic Field. It can do it not only in the role of an uninvolved observer, but also as a protagonist, identifying experientially with all the people, animals, plants, and even inorganic objects and processes that are part of this field" (Grov, p 19). Notable positive effects include oneness, ascertaining meaning, clarity of fear origins, closure, and integration of disturbing thoughts.

Accessing past lifetimes for the purpose of real time client healing in mental health settings has continued with others who further the validity and value of altered states work via past lifetime memories. Specifically, Dr. Brian Weiss, past life hypnotist and world renowned author of over a dozen books on past life transpersonal work, has demonstrated the benefits of past life integration in therapeutic settings. "Getting in touch with our past lives can profoundly and permanently heal [sic] mind and body" (Weiss, 2013). In his book: *Miracles Happen, The Transformational Healing Powers of Past Life Memories 2013*, Dr Weiss documents case studies where clients access their past lives in order to reconcile current lifetime emotional issues. In his book: *Many Lives, Many Masters 2021*, Dr Weiss transcribed what hypnotized clients described as "between lifetimes," or the waiting space of information, where one can observe and relay

objective information about their lifetime lessons. He documented that once client's remembered their past life trauma, they were able to better integrate the memory, assume a transcended state, and connect to the divinity and wholeness of their experience as a human being. (Weiss, 2013)

#### The Need for Akashic Research

Although the Akashic Record has been examined and described through science and used in case studies with prominent transpersonal healers for past life trauma integration, it has not yet been studied in a formal research design in a therapeutic setting. The Akasha has also not been used as an intervention tool in reducing mental health symptoms in any current or past research studies. The rising need of transpersonal interventions in therapy continues. Interest in spirituality is expanding. According to the Pew Research Center's Religious Landscape Study conducted in 2019, about 80% of U.S. adults say they believe in God or a higher power. Americans interested in increasing their spiritual growth jumped from 50% in the mid 1990's to over 80% in the twenty-first century" (Myers 2000). Furthermore, integrative approaches that involve altered state interventions such as holotropic breathwork, past life hypnosis, and psychedelic medicines are proving to be helpful in reducing mental health symptoms in clients.

With altered states work becoming more successful in mitigating negative symptoms, it is logical to increase research of other modalities within that framework to assess correlation. Especially modalities like the Akashic Records that are low risk, short in duration, produce immediate results, and pose little harm to clients. Transpersonal psychotherapy is a modality that seeks to establish a "conscious and growth-producing link between the patient and the transpersonal experience" (Canda and Smith, 2001, p.66). This growth-producing link, including the elements and impact, need to be further studied and defined in the context of negative symptom mitigation. Specifically, do Akashic Records sessions improve mental health outcomes as evidenced by a decrease in stress, anxiety, and depression, and/or an increase in resiliency and connectedness?

#### Study Design and Rationale

This study will be conducted in strict accordance with the ethical principles outlined in the Declaration of Helsinki (2013). Prior to the initiation of the study, ethics approval will be obtained from the appropriate institutional review board (IRB). Informed consent forms will be designed to prioritize the well-being, autonomy, and respect of all participants. The consent process will ensure that participants fully understand the nature, risks, and benefits of the study, and that their participation is entirely voluntary. Special consideration will be given to maintaining the privacy and confidentiality of participant information.

Our research will involve an analytical, experimental design with a transpersonal intervention of Akashic Sessions that involves past life records being read to participants by a licensed therapist who is trained in Akashic Records. Participants will complete 4, private, online, self-assessment evidenced-based rating scales before and after two Akashic sessions to measure baseline and post session mental health symptoms of anxiety, depression and stress. In addition, connectedness and resilience will be examined for coping and protective purposes. Participants will have two total Akashic sessions and some participants will engage in a semi-structured interview afterwards to gather qualitative data. The scales utilized will be: the

DASS Depression, Anxiety and Stress Scale, the WATTS Connectedness Scale, and the CD-RISC-10 Resiliency Scale.

The study design will mimic other low-risk, short, analytical and experimental research studies that employ a transpersonal intervention and seek to measure emotional or mental health symptoms using self-assessment rating scales. Specifically, the study: A Mindfulness-Based Intervention for Student Depression, Anxiety, and Stress: Randomized Controlled Trial by Ritvo et al, 2021, measured similar symptoms (anxiety and stress) and utilized self-assessment scales for stress and mindfulness that also included individual and group structured interviews to gather qualitative data. This study was also short-term where participants repeated scales to measure changes. In another study: An experience with Holotropic Breathwork is associated with improvement in non-judgement and satisfaction with life while reducing symptoms of stress in a Czech-speaking population by Uthaug et al, 2021, used an altered states intervention to examine stress by having participants complete 3 online self-assessment scales for multiple occurrences before and after a series of breathwork sessions to examine changes in mood and perception. Lastly, the study: Effectiveness of Transpersonal Therapy in Reducing Fear of Cancer Recurrence in Breast Cancer Survivors: A Randomized Controlled Trial by Sajadian, et al, 2021 employed transpersonal therapies such as yoga-meditation and spiritual discussion in therapy to examine fear levels in breast cancer patients. The method utilized was self-assessment scales for fear which were examined over the course of weekly interventions for several weeks and then analyzed. Within the scales, elements of resilience and coping were also noted.

# Summary

While transpersonal interventions have been increasing as a modern psychological tool, people are seeking meaning and spiritual engagement for emotional problems just as readily. "The best approach may involve the skillful combination of conventional psychotherapeutic techniques and the use of altered states transpersonal work" (Winter, 1999, p.18). While Akashic Records have been both validated by science and used in transpersonal work, its formal or measured application in mental health outcomes are sparse. The Akasha provides much potential for spiritual growth. For example, the ability to connect to deeper themes with trauma patterns, and to engage in depersonalization of internalized harmful beliefs are all consistent experiences for those having an Akashic Session. In essence, clients are moving outside of their current time-space reality, and engaging with their soul self. The benefits of Akashic Sessions are many, wherein the harm and risk are low.

With growing positive results for past life and altered states work to client wellbeing, and rising research for transpersonal interventions in simple, short-term, studies, it is both intuitive and logical to conclude that the Akasha is the next step along the road of a powerful trend in client healing modalities within transpersonal psychology.

#### 3. Inclusion and Exclusion Criteria:

#### Inclusion:

1. 18 years old and over

- 2. Ability and willingness to provide written, informed consent in English prior to initiation of any study-related procedures and adhere to all study requirements
- 3. Willingness to engage in discussion about past life patterns and emotions
- 4. Self report of anxiety, depressive or stress symptoms in the last 12 months

#### **Exclusion:**

- 1. Inability to provide consent due to cognitive impairment, mental health disorders, or other conditions that impact their ability to understand the nature, risks, and benefits of the study.
- 2. History of alcohol or substance use disorder within 12 months
- 3. History of hypomania or psychotic episode within 12 months
- 4. Prior history (lifetime diagnosis) of schizophrenia spectrum, or other psychotic disorders
- 5. Experiencing any other serious mental or physical health issues that would impact their ability to engage in the research study
- 6. Has either attempted suicide, has documented medical history of suicidal ideation, or been hospitalized due to suicide risk within 1 year prior to prescreening.
- 7. Previous Akashic Record Session with Interventionist, Candice S. Rasa, LCSW or previous Akashic Record Session with any other provider within 6 months.
- 8. Any form of medicinal therapy should be stable 3 months prior to screening with no plan to start, stop or alter the use of any prescribed medications, supplements or other therapies from informed consent
- 9. Any form of non-medical therapy should be stable 3 months prior to pre-screening with no plan to start, stop or alter use of psychotherapy, acupuncture, hypnosis, or other similar therapy from the time of providing informed consent.

# 4. Sample Size:

The anticipated total number of participants for this study is set at 100 individuals. This sample size is determined based on a careful consideration of several factors. 100 participants is often considered adequate for obtaining statistically significant results, particularly in studies with a single group (Mascha, 2018). This sample size strikes a balance between ensuring a sufficiently diverse representation of the population under investigation while also being manageable in terms of resources and time constraints. Additionally, the chosen sample size aligns with standard practices within the field and follows guidelines that recommend sample sizes to achieve statistical power (Brysbaert, 2019). A sample of 100 participants is generally

deemed suitable for detecting meaningful effects and relationships within the study's context. **Recruitment and Screening Methods:** 

**Recruitment Process:** The identification and recruitment of potential participants for the study will be conducted through a multifaceted approach. We will utilize exponential, discriminative snowball sampling, email recruitment, and public advertisement on the Rasa Healing, Inc. website and associated social media platforms.

All interested potential participants will be directed to a central landing page on the Rasa Healing Inc. website which objectively describes the study's purpose and inclusion and exclusion criteria. Potential participants will fill out a short online prescreen. Subsequently, our licensed clinician will conduct a pre-screening to determine eligibility. Any inquiries or concerns about the research will be directed to the research team.

Specifically, we will leverage the Rasa Healing email list via Flodesk by directly emailing subscribers of Rasa Healing Inc, providing them with information about the study and inviting them to review details on the landing page. Posts, graphics, and accompanying links to the landing page containing study details will also be made on the Rasa Healing Instagram account, Rasa Healing Facebook account, and Mighty Networks platform. Snowball sampling will also be employed, wherein clients of Candice Rasa and each participant of the research study will be asked if they recommend anyone else to participate.

# **5.** \*See Appendix D for Recruitment Materials

**Pre-Screening and Screening Process:** The screening process for participant eligibility in the study involves a multi-step approach utilizing online pre-screen questionnaire and pre-screen interviews. There will not be a separate informed consent provided for the pre-screening process and participants will not receive compensation for the pre-screening process. Initially, potential participants will be directed to a landing page containing detailed information about the study's purpose, procedures, and inclusion/exclusion criteria, with a link to a survey hosted on a HIPAA compliant platform, Jotform. Upon completion of the survey, participants will receive an automated email confirming their submission and provided a link to schedule a 30-minute virtual pre-screen interview via Google Meet, conducted by a licensed clinical social worker. Prescreening and post structured interviews will be conducted by a different licensed clinician than the one conducting Akashic Sessions.

During the pre-screen interview, the clinician will review the study procedures, timeline, and eligibility criteria with the participant and address any questions or concerns they may have. Participants will also be told why we are doing a screening process and what happens to the screening data for individuals who are not eligible to participate in the study. Eligibility will be assessed based on the outlined inclusion and exclusion criteria, with potential participants informed of their eligibility status during the call. Specific details as to why they do not qualify will not be provided to prevent attempts to alter responses. In cases where eligibility is unclear,

participants will be informed that they will receive a follow-up email or phone call once their status is confirmed, with the clinician consulting with the Principal Investigator regarding eligibility. All pre-screen questionnaires will be securely deleted from Jotform once it has been determined they are ineligible for the study.

If a participant meets the eligibility criteria, they will be provided with a copy of the informed consent form (ICF) and given the option to sign it electronically using Jotform during the pre-screen interview. Alternatively, participants may choose to review the ICF at their own pace and sign it electronically at a later time. They will be given the independent researchers' contact information to review any questions or concerns they may have at a later time prior to signing ICF. Upon signing the ICF and officially enrolling in the study, participants will be assigned a unique identification number to serve as their primary identifier throughout the study, ensuring confidentiality and data security.

\*See Appendix B for Prescreen script

\*See Appendix C for Prescreen checklist

#### 6. Research Locations:

Our study will be conducted solely online. We will use various online platforms for data collection, ensuring a comprehensive and efficient approach. Akashic sessions, Pre-screen interviews and semi-structured interviews will be conducted using Google Workspace. Within Google Workspace, we will use both Google Calendar for scheduling and Google Meet, a secure and reliable platform conducive to virtual interactions. In addition to Google Workspace, Jotform will serve as our primary platform for surveys, self-assessments, and questionnaires. Jotform is selected for its versatility and ease of use in creating, distributing, and collecting data from a wide range of forms. These platforms collectively offer a seamless and integrated online data collection process and are HIPAA compliant which will keep information stored securely.

For data collection from online sources, the study involves several preparatory steps to ensure compliance and confidentiality. Private visibility settings will be used for Google Calendar and utilized by authorized personnel with unique login credentials. This includes utilizing HIPAA compliant platforms, assigning private, password protected logins, de-identifying participant names, adding passwords to devices such as phones and computers used by the research team, and backing up data with an encrypted external drive. Measures such as confirming Business Associate Agreements with Google, internal staff training to limit PHI exposure, and maintaining audit logs, are implemented to ensure HIPAA compliance.

# 7. Multi-site Research (research that involves external collaborating institutions and individuals):

In addition to the primary investigator (Candice Rasa(, there are three independent contractors on staff who will serve as the co-investigator (Sarah Coleman), research coordinator (Betsy Koczab) and research staff (Briana Williams). Sarah Coleman, will function as the

co-investigator, and will be responsible for conducting pre-screen interviews with participants to assess their eligibility for the study. Following this, she will review each candidate with Candice Rasa to confirm eligibility. Sarah will review the informed consent form (ICF) with each participant, and obtain the signature of each participant who qualifies and wants to enroll in the study. Additionally, Sarah will provide guidance on navigating Google Meet and assist in scheduling appointments with Candice for the Akashic Record sessions. Furthermore, she will conduct semi-structured interviews with participants. Once the interviews are completed, she will analyze the collected data. Sarah will serve as the participant's primary point of contact for any questions or concerns they may have regarding the study.

Betsy Koczab, the research coordinator, her duties will encompass sending out emails and appointment reminders, participant communication regarding protocol procedures, timelines, and payments. Betsy will focus on the distribution of assessments or scales via email within the study timeline. She will also handle communication regarding rescheduling sessions, and confirming interviews are scheduled within the study timeline. Betsy will manage the distribution of session recordings to participants and uploading of session recordings onto an encrypted jump drive once a week. Betsy will also manage the study procedures and timelines for participants and staff.

Briana Williams, our research assistant, will also collaborate with the co-investigator to help analyze and code the semi-structured interviews. Together, they will contribute to the thorough analysis of the gathered data, ensuring comprehensive insights into the study's outcomes. Briana will not have access to participant interface, Google Workspace, Jotform, or any identifying client data. Briana will only have access to qualitative data de-identified, with UIN's, in the platform, Dedoose.

#### 8. Procedures Involved:

In this study, participants will undergo a series of research procedures, including self-report scales evaluating stress, anxiety, depression, resiliency, and connectedness before each of the two Akashic Records sessions and after the final session. The self-report scales include the CD-RISC-10 Connor Davidson Resilience Scale, DASS-21 Depression and Anxiety Scale, the Watt's Connectedness Scale, a demographic form and a brief satisfaction survey. The primary endpoint for this study is mental health and well-being which will be measured with the three self-report scales. The primary endpoint will be the third set of self-report scales that will be completed after the two Akashic Record sessions. Clients will complete surveys on their own, privately. The licensed clinician conducting Akashic Sessions will not have access to client feedback and surveys during the course of the study.

This study will not be accessing any secondary data sources, as they are not necessary to confirm eligibility or carry out our research objectives.

The primary research intervention involves two Akashic Records sessions facilitated by Candice Rasa, LCSW, a licensed clinical social worker, and certified Akashic Records channel. Each session, lasting approximately 50-90 minutes, will involve channeling the Akashic Record

for the participant, delving into areas such as past lives, emotional patterns, ancestral trends, and personally sensitive topics. Participants are encouraged to inquire about topics important to them, ensuring a personalized and participant-driven experience.

Akashic sessions will be scheduled on Google Calendar. A member of the research team will schedule the two Akashic sessions in advance with the participant after informed consent has been signed. Participants will also be taught how to reschedule or cancel their appointments on Google Meet and how to join their session online. [Please see Recording and Storage for more information on procedures involved for recording each Akashic session].

#### **Akashic Records Reader Methods**

Reading the Akasha involves a combination of intuitively receiving information from the Akashic field via psychic senses, using interpretation skills, translation of info to the participant via verbal dialogue, and holding space for the participant to respond and ask follow-up questions.

- Psychic senses used by readers are: empathy (psychic feeling), clairvoyance (psychic seeing/visualizing), clairaudience (psychic hearing), claircognizance (psychic knowing), and clairsentience (psychic sensing in the body).
- Interpretation skills are used by the reader to discern the information being received by the Akasha and this includes acknowledging the sense out loud to the participant. For example: "There is a feeling state of sadness being observed" or "A symbol of a flower is being shown and a phrase can be heard 'bloom.' The reader observes information received and relays it real time.
- Communication through verbal dialogue means relaying the information to the client in detail including past life storylines and deeper patterns associated with past life experiences. It also includes using skills such as linking, reflecting, summary, and clarification to connect themes together that arise from the introduction. Communication of Akashic themes is strictly focused on objective information-sharing versus clinical intervention.
- Participants are encouraged to speak openly and reflect on the themes and patterns presented and self-identify patterns, emotions, storylines, or themes that they wish to explore further by asking questions of the Akasha. Readers hold space for that by allowing participants self determination and asking transpersonal reflection questions.

#### **Akashic Record Channeling Verses Therapy:**

The Akashic Records is unique in its application and differs from therapy and coaching in key ways. Although therapy and Akashic Records may have shared intentions and outcomes, the methods for achieving client change are vastly different.

Therapy and Akashic Records are similar in that they may both be emotionally transformative, assist clients in understanding life problems from a new perspective, tease out strengths, or highlight self-defeating behaviors and thoughts, and alleviate negative symptoms associated with mental health diagnoses. Both modalities also involve private one on one exploration with a trained clinician with the intention of improving understanding and peace

about life circumstances through deeper self-exploration. Both modalities also pose a low risk for harm because the clients are self-determining topics discussed, are coherent and in sound mind and body, and are seeking/ are interested in talking about emotional themes.

However, perhaps the most notable difference between therapy and Akashic Records is the scope of how the clinician views the client and the source of information. While therapy does involve exploring past patterns and issues, Akashic Records considers these patterns from a transpersonal lens to include past lifetimes and ancestral themes that extend beyond the current time and space reality. This creates a much larger zoomed out perspective. In traditional therapy models, clients do not typically have a transpersonal experience, whereas in Akashic sessions clients regularly report sensations of deep seen-ness, connectedness, surrender, oneness and emotional release. Another major difference is the source of information that is discussed in session. While in therapy, clinicians derive client information from the client themselves, clinicians reading the Akashic Records source information from the Akashic field intuitively.

Several other differences are also noted. Therapy involves the therapist engaging in a mutual dialogue with the client, often talking less than the client in order to draw out client-led insights. Akashic Sessions are primarily information-sharing in nature where the client mostly listens and receives. Where therapy sessions are intended to help clients engage in introspection to discover insights about life patterns on their own, in Akashic channeling sessions, the reader offers the client insights about themselves based on past life records. In therapy sessions, clinicians analyze what the client is saying, redirects, reframes, and suggests interventions. In Akashic sessions, the reader responds only with psychological support and empathy.

#### **Akashic Records Procedure**

Akashic sessions include a specific session structure to assure consistency for each participant. Those components are:

- Prep discussion
- Channeled introduction
- Reflection period
- Q&A back and forth
- Summary and resource identification

#### Prep discussion

- All participants will receive the same prep sheet with general information on how to prepare for their session in advance. At least 1 week in advance.
- Session begins with preparation information on what to expect during the session including a review of what the Akashic Records are.
- See Appendix B for Akashic prep discussion script

#### Channeled introduction

• Akashic Records reader will read a short Akashic prayer aloud and encourage the participant to sit quietly for 2 minutes using slow deep breathing.

- Participants will be asked to reflect on the following: what is most important to them and what intention do they have for the session.
- Upon opening the Akashic Record with the specific prayer, the reader will then engage in an introduction; or spontaneous channeling of the participant's Akasha for approximately 5 to 10 minutes which includes past life and ancestral details and pattern identification. The participant sits quietly and receives this information.

## Reflection period

- Upon completion of the intro, the participant is encouraged to reflect, digest, and discuss any themes that arose for them upon listening to the introduction.
- The Akashic reader responds with psychological support. Psychological support is a non-directive approach and does not use a specific intervention or therapeutic modality like CBT or SFBT. Psychological support includes reflective listening and summarizing such as "what I heard you say was...", and statements that convey empathy. It may also include validation of the client's emotions or feelings. Creating a safe container in which the participant is given a non-judgemental and confidential space to share is also critical for providing psychological support.
- Statements of empathy and examples of psychological support may include the following:
  - o I am here for you
  - It is okay to cry and/or release
  - How would you like to be supported right now?
  - Take your time to gather your thoughts if you need them
- Akashic channel will trigger transpersonal reflection by asking the same process questions for each participant after channeled information is shared. Those questions are:
  - How is that landing for you?
  - How are you doing so far?
  - What's coming up for you?
  - How's that feeling in your heart?

#### Q&A back and forth

- The participant will be asked if there are specific questions or patterns that they would like to ask or know more about given their intention for the session and/or channeled introduction
  - What feels important for you to talk more about?
  - What questions do you have?
  - What's alive that you would like to talk about next?
  - Where would you like to go next?
- Participants will ask questions one at a time and Akashic reader will answer the questions by exclusively receiving information psychically from the Akashic field and relaying it as is to the participant.
- Patterns discussed include emotionally-focused exploration. Specifically, this means examining fears, emotions, and patterns around karmic and ancestral themes.

## Summary and resource identification

- Within 15 minutes of the session ending, the Akashic reader will review themes and patterns discussed in a summary and encourage additional questions or reflections about those topics from the participant
  - Is there anything more you wish to explore or ask more about?
- During the course of the session, if healing practices, resources, or suggestions were discussed, those are reviewed.
- Participant will be asked the following:
  - What is an important takeaway you would like to remember or reflect on further?
- When the Akashic Records are closed, the Akashic channel will read a completion script, see Appendix B

All Akashic sessions will be scheduled at mutually convenient times, recorded, and securely stored through a HIPAA-compliant database. While these recordings may be utilized for potential qualitative analysis, they will not be shared with anyone to maintain participant confidentiality.

Following the Akashic sessions, some participants will engage in a semi-structured interview approximately one week after their last reading. The research team will conduct structured interviews with participants with the aim of completing between 30 to 50 interviews. The decision to stop interviewing will be made collectively by the research team. This decision will be based on identifying redundancies in participant responses, indicating saturation of data. Regular meetings will be held to assess the progress of interviews and determine if additional interviews are necessary.

This interview, lasting approximately 1 hour, provides participants with an opportunity to elaborate on their experiences and discuss the perceived impact of Akashic Records sessions on their mental health.

It is important to note that no secondary data sources, such as student educational records or electronic health records, will be accessed for this study.

#### **Estimated Time Commitment**

The study will take approximately six hours of time across approximately three months (including the long-term follow-up). See timeline for further details:

#### **Phase 1: Application and Approval Process**

- o Initial Application: 10-20 minutes
- Pre-screen Interview: Approximately 1 hour
- Read and Sign paperwork: 10 minutes
  - Minimum 1 day prior to the first Akashic session. It must be completed before your session.

# Phase 2: Self Assessments and Akashic Readings

• First self-report assessment scales: 15 minutes

- Within 7 days of the 1st Akashic session. Must be completed before the session.
- Demographic Form
- CD-RISC-10 Connor Davidson Resilience Scale
- DASS-21 Depression and Anxiety Scale
- Watt's Connectedness Scale
- Initial Akashic Session: 90 minutes
  - No later than 30 days after pre-screen (or additional pre-screen will need to be conducted)
- Second set of self-report assessment scales: 15 minutes
  - Must be completed within 7 days of the second Akashic session. Must be completed prior to starting the second session.
  - CD-RISC-10 Connor Davidson Resilience Scale
  - DASS-21 Depression and Anxiety Scale
  - Watt's Connectedness Scale
- Second Akashic session: 50 minutes
  - 10-21 days after the first session

#### Phase 3: Final Assessments and Semi-Structured Interview

- Third set of self-report assessment scales: 15 minutes
  - 7-14 days after the 2nd Akashic session. Must be completed prior to semi-structured interview.
  - CD-RISC-10 Connor Davidson Resilience Scale
  - DASS-21 Depression and Anxiety Scale
  - Watt's Connectedness Scale
  - Satisfaction Survey
- o Potential Semi-Structured interview: Approximately 1 hour
  - 7 to 14 days after the final Akashic session
- Fourth set of self-report assessment scales: 15 minutes
  - 60 to 80 days after final Akashic session
  - CD-RISC-10 Connor Davidson Resilience Scale
  - DASS-21 Depression and Anxiety Scale
  - Watt's Connectedness Scale

#### **Self-Report Assessments**

Self-report scales will be completed on Jotform. Participants will be emailed a link to the corresponding forms and reminded of the timeframe they need to be completed by. Participants will be able to complete the self-report assessments privately and at their own pace. Participants will be reminded that Candice Rasa will not have access to seeing their self-report forms and that their information will remain confidential. We will use Jotform to analyze the quantitative data

from the self-report forms and analyze the changes in the scores based on pre and post Akashic sessions.

## **Semi-Structured Interview**

While not all participants will partake in the semi-structured interview, our team aims to interview the first 30 to 50 individuals in the study. This target range was chosen based on previous research on qualitative analysis, identifying the optimal number of interviews to ensure comprehensive data collection. The research team will meet regularly to discuss data saturation, meaning that new insights and themes cease to emerge, indicating that a thorough exploration of the topic has been achieved without excessive redundancy.

This range of participants for a semi-structured interview in a qualitative study is considered appropriate for several reasons. This number allows for a diverse range of perspectives and experiences to be captured, ensuring a comprehensive understanding of the research topic. It also provides sufficient depth in the data collected, allowing for proper analysis and interpretation. Finally, managing a sample size within this range is practical in terms of time, resources, and the feasibility of conducting in-depth interviews while maintaining rigor in data collection and analysis.

Interviews will be scheduled with the independent evaluator who is a licensed clinical social worker. Interviews will be completed about one week after the second Akashic Record session. Participants will be able to sign up for a timeslot on Google Meet and they will be automatically sent the meeting time and date as well as a link to access the virtual meeting.

During the interview, the interviewer will read a script which provides information on why and how the interview is being conducted. Participants will be reminded that the interviews are recorded and that their information will remain confidential. Participants will be informed that they can ask to stop the recording at any time. The interviewer will use questions as a basic guideline for the interview and use reflective listening and follow-up questions to get detailed information regarding their experiences with the Akashic sessions.

Interviews will then be transcribed verbatim into Jotform by the independent evaluator. Once the interviews are transcribed, they will be reviewed and coded using a secure HIPAA compliant software called Dedoose which allows for data storage and analysis. We will look for repeating themes and categories throughout each interview and code them based on the recurring themes. To ensure consistency and rigor in our coding process, we will implement interrater reliability measures. Specifically, two individuals will independently code the interviews and engage in regular discussions to reconcile any discrepancies and ensure alignment of viewpoints. This collaborative approach will enhance the validity and reliability of our qualitative data analysis. Once each interview is coded, we will analyze and draw conclusions based on how the different themes relate to one another and how they relate to the self-report changes in scores.

\*See Appendix B for Semi-Structured Interview Script

#### **Participation**

1. What motivated you to seek help through the Akashic Record sessions? [Areas for probing: What did you want to improve or work on? What were you hoping or expecting to get out of these Sessions?]

#### The Akasha

2. Did you know about the Akasha before joining in this study? [Areas for probing: Can you share more about how your understanding of the Akasha has changed over the course of the 2 sessions provided?]

#### **Benefits**

- 3. Thinking back on your experiences, what parts of the sessions did you find most helpful?
- 4. Can you share about your view of your challenges or problems compared to before you started this study? [Areas for probing: Can you share any specific insights you gained during the sessions that helped you in working on your challenges?]

# **Integration**

- 5. How has the process been for you since your second session? How has it been integrating the new insights that you got from the sessions into your daily life?
- 6. Can you share whether you used the interventions or practices that were suggested to you during your session? Why or why not?

# **Challenges**

7. Were there any other difficulties you faced during or after the sessions? If so, can you share some details about those experiences?

# 9. Research with Vulnerable Populations

While we are not purposefully recruiting participants from groups formally designated as "vulnerable populations," we will also not deny someone inclusion in this study because of a self identified vulnerability status, i.e., pregnant women, persons with disabilities, etc.

# 10. Incomplete Disclosure or Deception:

N/A

#### 11. Consent Process:

The consent process for our study will be conducted at the end of the virtual pre-screen interview by a licensed clinical social worker. Participants will have the purpose, timeline, and confidentiality details of the study explained to them verbally. They will have the opportunity to ask questions, and a copy of the informed consent will be emailed to them for review and signature. The Co-PI/ licensed clinical social worker/ independent evaluator Sarah Coleman, LCSW will be a witness when the participant signs the ICF. She will sign the form after they have completed it. The informed consent will be written in clear simple terms to ensure participants fully understand what it means to participate in the study. Participants will be reminded throughout the study that it is in their right to withdraw from the study at any time and that there will be no consequences or repercussions. The signed consent form will be documented, and participants will find contact information on the form for any additional questions or concerns. This process ensures participants understand the research procedures and can make an informed, voluntary, decision to participate.

Further details on the consent process is outlined in Appendix A, Standard Operating Procedures

# 12. Research with Children – Parental Permission, Child Assent, and Other Considerations:

N/A

# 13. Waiver of Participant Signature on Consent Form:

We are not allowing the option of waving signatures on consent forms. If someone is not cognitively or physically capable of providing informed consent, they will not be included in the study.

#### 14. Waivers and Alterations of Consent Information:

N/A

# 15. Financial Compensation:

There is no monetary compensation for participating in this research. However, participants will receive a discount of 15% off each Akashic Records session. The intake session is 90 minutes and \$379 (research participants will pay \$322), follow-up sessions are 50 minutes at the rate of \$239 per session (research participants will pay \$203). In total, new participants will save \$93 across the two sessions. Participants will be billed prior to each Akashic Session.

Participants will be charged for sessions to maintain consistency with real-world Akashic sessions. This allows for research variables to stay consistent and acknowledges the presence of a financial investment that, in a typical setting, may correlate with increased commitment levels. Compensation in the form of a discount is offered to account for the additional time and effort it may take for participants to complete study self report assessments.

There will not be extra costs to subjects or third-party payers for their participation in the study.

# 16. Audio/Video Recording/Photography:

The research study employs a recording process integral to the research methodology, capturing essential data for analysis and to replicate real world scenarios for participants. Recordings of both Akashic Sessions and semi structured interviews are securely stored and managed following strict protocols to safeguard participant confidentiality and comply with HIPAA regulations.

For Akashic Record sessions, recordings are captured via Google Meet, a confidential platform compliant with HIPAA regulations. The recording process is initiated once a verbal confirmation is given by the participant at the beginning of the Akashic Session and they have confirmed they are comfortable discussing personal information and they are in a confidential and private space. The purpose of recording Akashic Sessions is to mimic real world sessions so that participants can receive and relisten to their Akashic Sessions, which supports integration and revisitation of session concepts. For Akashic Sessions, the Research Coordinator will send session recordings to participants via Google Workspace secure email link. For added privacy, links to session recordings will only be authorized to the password protected email associated with the participant.

In addition to Akashic Record sessions, semi structured interviews are also recorded via Google Meet as part of the research methodology. These recordings capture participant responses and interactions during structured interviews. The recording process for interviews ensures the preservation of participant input, facilitating detailed analysis and interpretation of data. The recording process is initiated once a verbal confirmation is given by the participant at the beginning of the interview and they have confirmed they are comfortable discussing personal information and they are in a confidential and private space.

Following both Akashic sessions and semistructured interviews, recordings are automatically transferred to a designated, password-protected cloud storage within Google Workspace's Drive available only to credentialed research staff with unique logins. Specifically, recordings will be stored in a password protected folder in Google Drive, which Candice Rasa will not have permission to access. Duplicate copies of the recordings will be made on encrypted, password enabled, jump drive for additional security. Access to these recordings is restricted to authorized personnel within the research team, who adhere, and are trained, in HIPAA compliance standards. The original recordings will be permanently deleted from Google Workspace platforms to uphold participant confidentiality. It is important to note that while voices and information will be recorded during the sessions, no names or identifying information will be included to protect participant anonymity. All recordings are retained for a period of 6 years. Any incidents of unauthorized access or breaches are promptly reported to the IRB and relevant authorities with appropriate measures taken to address and mitigate such incidents.

## 17. Potential Benefits of this Research:

Akashic Record sessions offer participants the potential for a resolution of personal issues, as insights and perspectives gained during the sessions can be impactful. These sessions

may provide participants with a clearer understanding of unresolved emotional issues, offering newfound awareness of how to address these matters. Moreover, the sessions may trigger realizations of hidden strengths within participants, empowering them to navigate challenges with a deeper understanding of their capabilities and confidence in themselves. Accessing the Akashic records can further activate participants' resiliency, enabling them to cope more effectively with life's challenges and setbacks. This may include improvements in mood and emotional coping due to altered state consciousness and connection to a larger why. Additionally, the exploration of the Akashic records may lead to a profound sense of peace, purpose, and meaning in participants' lives.

The research on Akashic Record sessions not only holds the promise of enhancing individual well-being through personal growth and improved emotional well-being but also suggests potential societal benefits. The activation of resiliency at the individual level could extend to communities, fostering increased collective resilience and an improved ability to overcome adversity. Additionally, participants gaining insights into their emotions and behaviors may contribute to the cultivation of healthier interpersonal relationships, positively influencing the social fabric.

# 18. Risks to Participants:

Akashic Records sessions involve relaying information to clients about past lifetimes, ancestral patterns, and karmic relationships. These sessions can be intensely personal and bring up undesired strong emotions. Participants may experience discomfort in completing self-assessment rating scales and/or be unable to complete surveys within study parameters. Participants may not be able to meet for Akashic Record sessions due to work, family and/or other personal or life responsibilities. Participants may not want to share honestly or openly in surveys due to fear of giving negative feedback to Akashic Records clinician. Participants may not know how to navigate the digital platforms where the surveys are housed. Participants may fear their private information will be shared with others. Participants may not be able to afford Akashic Sessions as part of the study, so paying for sessions may cause distress. While these are all potential risks, past Akashic Records clients have reported that the sessions have highly positive outcomes rather than negative, and engaging in Akashic Records sessions greatly enhances and expedites therapeutic process.

In order to minimize emotional risk and client harm there are licensed clinicians as a part of the study team. All Akashic Records sessions will be conducted by a licensed clinician with over 15 year's experience and training in transpersonal methods including Akashic channeling. The Akashic interventionist has active experience in seeing 15 to 20 clients weekly for Akashic Sessions in the last 6 years as part of an existing practice and is familiar with diverse clients, procedures, and in managing a variety of client responses. Psychological support will also be offered as needed during sessions. The independent evaluator who will be supporting participants throughout the research study is also a licensed clinician and will be able to connect participants to additional resources when needed. As part of the study process, participants will be given a referral list (see Appendix for more details) with different mental health resources as part of the study completion procedures. If they need additional support, they will be connected to services immediately during or after the study.

As part of the exclusion criteria, clients will be screened out for active suicidal ideation, active thought-disorder, psychotic diagnoses or symptomology, and active substance abuse or dependence. Participants with these diagnoses will be excluded from the study to minimize psychological distress. A referral list will be developed and offered to any client in any part of the research process who is presenting, needing, or requesting additional mental health referrals. This includes prescreen clients not yet admitted into the study, accepted participants, post study clients at the end of the study. Participants will be informed that they can exit the study at any time they wish.

Breach of confidentiality is a potential risk. To mitigate this risk, a user friendly, HIPAA compliant, platforms have been purchased (Jot Form, Google Meet, Dedoose) to keep participant information confidential and to house surveys and data in an organized, protected way. Our pre-screen process will include a tutorial in using the digital platform for participants. No session recordings will occur without verbal consent of participants. The PI and Co-PI are licensed clinicians and therefore trained in HIPAA compliance, bound by the NASW code of ethics, and Florida law to maintain confidentiality. The research team is trained in HIPAA compliance. Password protection, encryption, and participation de-identification will be utilized

# 19. Provisions to Protect Participant Privacy and Data Confidentiality:

# **Participant Privacy:**

**Recordings**. Participants will be explicitly informed about the recording process during the informed consent phase, and their explicit consent will be obtained before initiating any assessment form, Akashic session, or recording. The recordings of the Akashic record sessions and interviews will be securely stored in an encrypted jump drive and a password protected server on Google Workspace with restricted access to the research team only. Any identifiable information shared during the recorded sessions, including personal details or specific experiences, will be carefully redacted or anonymized in the recordings to ensure confidentiality. The research team will emphasize the importance of using these recordings solely for research purposes.

**Physical environment.** During the Akashic record sessions and the semi structured interview, careful consideration will be given to the physical environment to ensure privacy. Each session and interview will be conducted in private spaces, where the conversations cannot be overheard by others. The interviewer will ask participants before starting the interview if they are in a place where they feel comfortable sharing confidential information. This helps create a confidential setting, allowing participants to openly share their experiences without concerns about the information being disclosed to unauthorized individuals.

**Storage**. Participants will be informed about the secure storage of data, de identification of personal information, and the restricted access to personal information. Additionally, they will have the opportunity to specify any preferences or limitations regarding the handling of their data. Client information will only be stored in HIPAA compliant, password protected, digital platforms and accessed only by authorized personnel relevant to their role in the study. No client information or research data will live outside of Google Workspace, Jotform and Dedooze and

unique identification numbers will be assigned to participant data to minimize confidentiality leaks.

# **Confidentiality of data/biospecimens:**

There will be no collection of any biospecimens for this study. For data collection, once participants have signed the informed consent form and officially joined the study, they will receive a unique identification number (UIN), beginning with "0001" and increasing sequentially with each new participant enrolled. These numbers, along with participants' names, will be recorded in a spreadsheet on Google Workspace for reference.

The online project management platform Monday.com will be used to manage adherence to study timelines for each participant. Only UIN's will be listed alongside study timeline checklists. Monday.com is a HIPAA compliant platform and only research staff will have access via password only access. No client names or identifiable data will be listed here. Throughout the study, the UIN will serve as the primary identifier for each participant, utilized in all storage of recorded data, including Akashic session recordings and interviews and qualitative data, ensuring consistency across all platforms and documentation.

To maintain compliance with HIPAA regulations and data security standards, procedures will be regularly reviewed and updated, with access to participant data restricted to authorized personnel only, and strict confidentiality and secure storage protocols upheld. Periodic reviews and updates of the Standard Operating Procedure (SOP) will be conducted to reflect any changes in procedures or regulations, with staff involved in participant enrollment and data management receiving training to ensure adherence to the SOP and HIPAA compliance.

# **20.** Data Monitoring Plan to Ensure the Safety of Participants:

The Research Coordinator will be responsible for the following tasks as part of data monitoring for continuity and participant safety:

- Conduct weekly audits of data protection procedures
- Be responsible for communicating with participants for self assessments and study timeline adherence for confidentiality and ease of process.
- Ensure procedural compliance of staff checklists and follow through on confidentiality protocols via weekly research team meeting
- Monitor conflict of interest and maintain passwords to Jotform so that Candice Rasa, will not have access
- Upload recordings to secure encrypted drive
- De-identify participant data. Specifically, ensure UIN's are listed on project management platform and for all recordings of Akashic Sessions and semi structured interviews
- Regularly review research protocol and procedures for compliance
- Co-responsible for reporting adverse events and/or breaches of confidentiality with independent evaluator to IRB and associated required bodies

# 21. Long-term Data and Specimen Storage and Sharing:

Recordings stored on encrypted jump drives, and data from the survey results as well as transcripts from the semi-structured interviews will remain in the password protected and HIPAA compliant website Jotform. This data will be stored in Jotform and the encrypted jump drive for a 6-year retention period and used for potential future research with inactive participants. The data may be moved into a reputable database upon approval of additional studies. The selection of a database will be contingent upon factors such as the adherence to data security standards, accessibility, and compatibility with the nature of the research data. Identifiers will not be included with the shared data to uphold participant confidentiality and privacy, consistent with ethical research practices. This approach underscores our commitment to safeguarding participant anonymity and ensuring responsible data management throughout the research.

# 22. Qualifications of Research Team to Conduct the Research:

**Principal Investigator and Sponsor:** Candice Rasa, LCSW is the Founder of Rasa Healing and has 17 years' experience utilizing transpersonal, existential, and humanistic therapy to catapult soul-level transformation in clients. Candice earned a bachelor's degree, Magna cum laude, in 2003 in legal studies with a minor in psychological studies from Nova Southeastern University. Candice earned a Master's in Clinical Social Work, Summa cum laude, in 2005, from Florida International University. Candice has been a licensed clinical social worker since 2007 and state of Florida Qualified Supervisor since 2009.

Candice was trained in Akashic Records at the Divine Love Institute in 2012 and completed certification of the highest available course: Advanced Akashic Records reading. Candice also completed psychic development certification in the Sandy Anastasi system of psychic development in 2015. Candice has been reading the Akashic Records in her current private practice for 9 years. Candice sees an average of 18 clients a week exclusively for Akashic Records readings and integrative therapy. Candice also completed karma yoga at the Kripalu Center for Yoga and Health and is certified in Integrated Energy Therapy, JourneyDance, Channeling/Mediumship and mindfulness meditation techniques. Candice regularly guest teaches at FAU and Lynn University on the value of alternative and complementary spiritual therapies and presents at the Florida National Association of Social Work conference annually on transpersonal clinical interventions.

Candice completed NIDA Good Clinical Practice Certificate and the CITI Program Human Subjects Research Certificate. Candie also has several CEU's on ethics, boundaries and HIPAA compliance since licensure in 2007 (see CV for more).

**Co-Investigator and Independent Evaluator:** Sarah Coleman, LCSW has her Masters of Social Work from Florida International University and a Bachelor of Social Work from the University of Illinois at Urbana Champaign. She has been working in mental health for over five years.

Sarah has worked in clinical research at Segal Trials since August 2022 as both a Screening Specialist and a Psychedelic Therapist. She has been trained and worked as a

co-facilitator for psychedelic dosing sessions and provides preparation and integration sessions. Sarah also has experience with reviewing and training staff members on study protocols and assisted in the screening process by assessing participant eligibility based on study protocols. Sarah has previous experience working on a study which explored the barriers to treatment for women with opioid use disorder. Sarah worked alongside an assistant professor at FIU helping conduct, code and transcribe interviews with women with opioid dependency.

Sarah completed CITI Biomedical Research Certificate, CITI COI Certificate, CITI Good Clinical Practice (GCP) Certificate, and a CSSRS Certificate. She also is trained in internal staff HIPAA compliance procedures and Research protocols workflow.

**Research Coordinator:** Betsy Koczab has a versatile skill set across various domains, notably as an Executive Assistant and Project Manager. She has experience managing sensitive information, and ensuring confidentiality for high-profile executives. while navigating complex administrative landscapes.

As a Project Manager, she engages directly with clients, facilitating seamless communication and collaboration. She has experience coordinating virtual meetings,managing projects across different industries and task delegation. Betsy's journey also extends to supporting professionals in mental health settings, where she plays a crucial role in managing administrative tasks with sensitivity and care. This includes handling confidential client information and maintaining privacy standards in therapy sessions, exemplifying her commitment to ethical practices. Betsy's diverse background has provided a solid theoretical foundation in research methodologies, ethics, and data management.

Betsy has received certifications from the CITI Clinical Research Coordinator (CRC) training and NIDA Good Clinical Practice (GCP) training. She also is trained in internal staff HIPAA compliance procedures and Research protocols workflow.

Research staff/ Data analyst: Briana's diverse skill set and extensive experience qualify her as an excellent research assistant. She is proficient in handling sensitive client information and utilizes HIPAA-compliant tools like Practice Better. Additionally, Briana has in-depth knowledge of various web analysis tools, including Omniture Site Catalyst, Test & Target, Webrends, Maxymizer, Tealeaf, and Foresee Results. She has utilized these tools to provide valuable insights to stakeholders through both qualitative and quantitative data analysis spanning over eight years. Briana meticulously orchestrated the test design for A/B and multivariate experiments on prominent corporate websites, ensuring randomized controlled testing procedures were flawlessly executed. Following data collection, she conducted thorough analyses, delving into various sub-populations to discern nuanced differences in outcomes based on demographic or behavioral variations within the audience.

Briana has also successfully managed both local and offshore teams to improve data reliability and validation while ensuring timely project completion. She excels in communicating

findings to stakeholders, even in challenging situations, and has led cross-functional teams to enhance user experiences based on data insights. Briana is committed to excellence and consistently seeks ways to streamline processes and enhance user design.

Briana is also trained in internal staff HIPAA compliance procedures and in Dedoose tutorials for data analyzation specialization.

#### 23. References

Álvarez-García, C., & Şimşek Yaban, Z. (2020). The effects of preoperative guided imagery interventions on preoperative anxiety and postoperative pain: A meta-analysis. *Complementary Therapies in Clinical Practice*, 38, 101077. <a href="https://doi.org/10.1016/j.ctcp.2019.101077">https://doi.org/10.1016/j.ctcp.2019.101077</a>

Bache, C. M. (2006). Reincarnation and the Akashic field: A dialogue with Ervin Laszlo. *World Futures*, 62, 114–126. https://doi.org/10.1080/02604020500406109

Blavatsky, H. P., & Horne, A. (2013). Alchemy and the secret doctrine. Literary Licensing.

Brysbaert, M. (2019). How many participants do we have to include in properly powered experiments? A tutorial of power analysis with reference tables. *Journal of Cognition*, 2(1), 16. <a href="https://doi.org/10.5334/joc.72">https://doi.org/10.5334/joc.72</a>

Buckley, P., & Galanter, M. (1979). Altered states of consciousness during psychotherapy: Historical and cultural perspectives. *International Journal of Social Psychiatry*, *25*(2), 118–124. https://doi.org/10.1177/002076407902500203

Camelo, L. G. (2022). The role of consciousness in healing therapies: A brief history of ancestral energies, biofield and ultra-weak photon emission. *Open Journal of Medical Psychology, 11*(2), 39–56. <a href="https://doi.org/10.4236/ojmp.2022.112004">https://doi.org/10.4236/ojmp.2022.112004</a>

Canda, E. R. (2012). Spirituality in social work. Routledge.

Canda, E. R., & Smith, E. D. (2001). *Transpersonal perspectives on spirituality in social work.* Haworth Press.

Chidambaram, A. G., & Josephson, M. (2019). Clinical research study designs: The essentials. *Pediatric Investigation*, *3*(4), 245–252. <a href="https://doi.org/10.1002/ped4.12166">https://doi.org/10.1002/ped4.12166</a>

Chow, W. M., Wooten, H. R., & Leonard, H. T. (2008). Breathwork and couple relationships: A qualitative investigation. *Journal of Heart-Centered Therapies*, 11(1), 91–112.

Collins, M. (2011). The Akashic field and archetypal occupations: Transforming human potential through doing and being. *The Journal of Global Education*, *67*, 453–479.

Frankl, V. E. (1946). Man's search for meaning. Beacon Press.

Grof, S. (2006). Ervin Laszlo's Akashic field and the dilemmas of modern consciousness research. *World Futures*, 62(1–2), 86–102. https://doi.org/10.1080/02604020500406091

Grof, S. (2008). Brief history of transpersonal psychology. *International Journal of Transpersonal Studies*, 27(1), 46–54. https://doi.org/10.24972/ijts.2008.27.1.46

Hertzog, M. A. (2008). Considerations in determining sample size for pilot studies. *Research in Nursing & Health*, 31(2), 180–191. https://doi.org/10.1002/nur.20247

Jonas, W. B., & Crawford, C. C. (2003). Healing, intention and energy medicine: Science, research methods and clinical implications. Elsevier.

Jung, C. G. (2001). *Modern man in search of a soul* (W. Dell & C. Baynes, Trans.). Routledge Classics.

Kaspersen, M., & Hårklau, H. (2008). Emotional processing: Psychotherapy and altered states of consciousness—Principles, therapeutic possibilities and challenges. *Psykologisk Tidsskrift, 3,* 19–25.

Kasprow, M. C., & Scotton, B. W. (1999). A review of transpersonal theory and its application to the practice of psychotherapy. *Psychotherapy Practice*, 8(1), 12–23.

Keppler, J. (2021). Building blocks for the development of a self-consistent electromagnetic field theory of consciousness. *Frontiers in Psychology, 12*, 850572. https://doi.org/10.3389/fpsyg.2021.850572

Krippner, S. (2006). Geomagnetic field effects in anomalous dreams and the Akashic field. *World Futures*, 62(1–2), 103–113. https://doi.org/10.1080/02604020500406117

Lajoie, D., & Shapiro, S. (1992). Definition of transpersonal psychology: The first twenty-five years. *Journal of Transpersonal Psychology*, 24, 79–98.

Laszlo, E. (2007). Science and the Akashic field: An integral theory of everything. Inner Traditions.

Laszlo, E. (2014). *The self-actualizing cosmos: The Akasha revolution in science and human consciousness.* Inner Traditions.

Levin, J. (2019). Western esoteric healing II: A taxonomy of sources of therapeutic knowledge. *Explore*, 17(2), 153–161. https://doi.org/10.1016/j.explore.2018.11.003

Levin, J. (2020). Hacking the Akashic records: The next domain for military intelligence operations? *Journal of New Paradigm Research*, *76*(2), 102–117. https://doi.org/10.1080/13537903.2020.1740203

Mackey, L. J. (2007). The collective unconscious and the Akashic field. *Jung Journal: Culture and Psyche*, *I*(2), 2–15. https://doi.org/10.1525/jung.2007.1.2.2

Mascha, E. J., & Vetter, T. R. (2018). Significance, errors, power, and sample size: The blocking and tackling of statistics. *Anesthesia & Analgesia*, 126(2), 691–698. https://doi.org/10.1213/ANE.0000000000002741

Matos, L. C., Machado, J. P., Monteiro, F. J., & Greten, H. J. (2021). Perspectives, measurability and effects of non-contact biofield-based practices: A narrative review of quantitative research. *International Journal of Environmental Research and Public Health*, *18*(12), 6397. <a href="https://doi.org/10.3390/ijerph18126397">https://doi.org/10.3390/ijerph18126397</a>

Miller, T., & Nielsen, L. (2015). Measure of significance of Holotropic Breathwork in the development of self-awareness. *Journal of Alternative and Complementary Medicine*, *21*(12), 793–803. https://doi.org/10.1089/acm.2015.0084

Nash, A. (2019). The Akashic records: Origins and relation to Western concepts. *Central European Journal of Contemporary Religion*, *2*, 109–124. https://doi.org/10.14712/25704893.2019.6

Pascual-Leone, A. (2016). The client "experiencing" scale as a predictor of treatment outcomes: A meta-analysis on psychotherapy process. *Psychotherapy Research*, 27(6), 1–13.

Pascual-Leone, A., & Yeryomenko, N. (2017). The client "experiencing" scale as a predictor of treatment outcomes: A meta-analysis on psychotherapy process. *Psychotherapy Research*, 27(6), 653–665. <a href="https://doi.org/10.1080/10503307.2016.1152409">https://doi.org/10.1080/10503307.2016.1152409</a>

Plante, T. G. (2008). What do the spiritual and religious traditions offer the practicing psychologist? *Pastoral Psychology*, *56*, 429–444. https://doi.org/10.1007/s11089-008-0123-6

Romney, A. K., Weller, S. C., & Batchelder, W. H. (1986). Culture as consensus: A theory of culture and informant accuracy. *American Anthropologist*, 88(2), 313–338. https://doi.org/10.1525/aa.1986.88.2.02a00020

Rubik, B. (2015). Biofield science and healing: History, terminology, and conceptual foundations. *Global Advances in Health and Medicine*, *4*(Suppl), 8–14. <a href="https://doi.org/10.7453/gahmj.2015.038.suppl">https://doi.org/10.7453/gahmj.2015.038.suppl</a>

Sagi, M. (2022). The role of information in classical and modern paradigms. *Journal of New Paradigm Research*, 7(3), 386–393. https://doi.org/10.1080/13537903.2022.2106340

Sajadian, A., Zahrakar, K., & Asadpour, E. (2021). Effectiveness of transpersonal therapy (spiritual therapy, yoga-meditation) in reducing fear of cancer recurrence in breast cancer survivors: A randomized controlled study. *Iranian Quarterly Journal of Breast Disease*, 14(2), 85–97.

Sheldrake, R. (1987). Mind, memory, and archetype: Morphic resonance and the collective unconscious—Part I. *Psychological Perspectives*, *18*(1), 9–25. https://doi.org/10.1080/00332925.1987.10559258 Siegel, D. J. (2023). Toward an interpersonal neurobiology of awareness: The probability position and the plane of possibility. *Frontiers in Psychology, 14,* 989760. https://doi.org/10.3389/fpsyg.2023.989760

Siegel, I. R. (2013). Therapist as a container for spiritual resonance and client transformation in transpersonal psychotherapy: An exploratory heuristic study. *Journal of Transpersonal Psychology*, 45(1), 49–74.

Steiner, R. (1987). Cosmic memory. SteinerBooks.

Tart, C. T. (1990). Altered states of consciousness. Harper.

Todeschi, K. J. (1998). Edgar Cayce on the Akashic records: The book of life. A.R.E. Press.

Uthaug, M. V., Lancelotta, R., Szabo, A., Davis, A. K., Riba, J., & Ramaekers, J. G. (2019). Prospective examination of synthetic 5-methoxy-N,N-dimethyltryptamine inhalation: Effects on salivary IL-6, cortisol levels, affect, and non-judgment. *Psychopharmacology*, *237*(3), 773–785. <a href="https://doi.org/10.1007/s00213-019-05414-w">https://doi.org/10.1007/s00213-019-05414-w</a>

Uthaug, M. V., Mason, N. L., Havenith, M. N., Vancura, M., & Ramaekers, J. G. (2021). An experience with Holotropic Breathwork is associated with improvement in non-judgement and satisfaction with life while reducing symptoms of stress in a Czech-speaking population. *Journal of Psychedelic Studies*, *5*(3), 176–189. https://doi.org/10.1556/2054.2021.00158

Watjen, L. (2014). An argument for the use of Holotropic Breathwork as an adjunct to psychotherapy. *Journal of Transpersonal Research*, 6(1), 103–111.

Weide, T. N. (n.d.). Varieties of transpersonal therapy. In *Journal of Transpersonal Research* (pp. 7–15).

Weiss, B. (1994). Many lives, many masters. Piatkus.

Weiss, B. L., & Weiss, A. E. (2012). Miracles happen. Harper Collins.

Zemła, K., Postępski, F., Kwaśniewicz, Ł., Kawiak, A., & Wójcik, G. M. (2023). Investigating the impact of guided imagery on stress, brain functions, and attention: A randomized trial. *Sensors*, *23*(13), 6210. <a href="https://doi.org/10.3390/s23136210">https://doi.org/10.3390/s23136210</a>

#### APPENDIX A

#### **Procedures**

i. Title: Procedure for Participant Identification and Recruitment

Version: [1]

Effective Date: [5.8.24] Review Date: [5.8.24]

**Objective:** To outline the process for participant identification in recruitment and marketing for the Akashic Record Research Study in accordance with Institutional Review Board (IRB) guidelines, ensuring compliance with ethical standards and participant safety.

**Scope:** This procedure includes all those involved in the recruitment and marketing process.

## 1. Identifying Potential Participants:

- 1.2 Potential participants will be identified through a combination of strategies including exponential, discriminative snowball sampling, and public advertisement on platforms associated with Rasa Healing, Inc.
- 1.3 The research team will leverage the Rasa Healing email list to reach out to adults directly via email using publicly available contact information.

#### 2. Invitation to Participate:

- 2.1 Invitations to participate will be extended through various channels, primarily targeting individuals interested in mental health and holistic healing.
- 2.2 Recruitment efforts will include publishing professional and objective posts on social media platforms such as Rasa Healing's Instagram account, providing a brief overview of the study's purpose and general inclusion/exclusion criteria.

#### 3. Recruitment Strategies and Materials:

- 3.1 Online Platforms: Utilization of online recruitment strategies will involve posting recruitment information on Rasa Healing, Inc.'s website and social media pages, including Instagram, Facebook, and Mighty Network professional pages.
- 3.2 Email Campaigns: A landing page detailing study information will be shared via Flodesk email platform with all subscribers of Rasa Healing, Inc. Additionally, an email template containing study details will be sent to subscribers.
- 3.3 Snowball Sampling: Participants of the study and clients of Candice Rasa will be asked to recommend individuals for potential participation, thereby initiating a snowball sampling approach.

# 4. Application Process:

- 4.1 All individuals interested in participating in the research will be required to fill out a short online application providing basic contact information.
- 4.2 The online application will serve as an initial expression of interest from potential participants.

#### 5. Pre-Screening and Eligibility Determination:

- 5.1 A licensed clinician from the research team will conduct a pre-screening via phone to determine the eligibility of potential participants based on predetermined criteria.
- 5.2 Direct contact will be made with potential participants to assess their suitability for inclusion in the study.

#### 6. Handling Inquiries:

6.1 Any questions or comments about the research will be directed to the research team, who will promptly address inquiries and provide necessary information to interested individuals.

## 7. Marketing Tools and Locations:

- 7.1 The study details, including purpose and inclusion/exclusion criteria, will be prominently displayed on a landing page on Rasa Healing, Inc.'s website.
- 7.2 Graphics containing study information will be posted on Rasa Healing's social media platforms, with accompanying links to the landing page for further details.

# 8. Compliance and Review:

- 8.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 8.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 8.3 Research team will meet weekly to review study procedures, timeline. And compliance.

# ii. Title: Standard Operating Procedure for Participant Eligibility Confirmation


Effective Date: [5.8.24] Review Date: [5.8.24]

**Objective:** To confirm the eligibility of participants in the Akashic Record Research Study in accordance with Institutional Review Board (IRB) guidelines, ensuring compliance with ethical standards and participant safety.

**Scope:** This procedure includes all those involved in eligibility determination and enrollment and specifically, PI and Co-PI

### 1. Landing Page and Survey:

- 1.1 Potential participants will be sent a landing page which has a detailed description of the study's purpose, procedures, and basic inclusion/exclusion criteria as well as a link to a survey hosted on a HIPAA compliant Jotform platform.
- 1.2 Potential participants will then be directed to complete a short survey with questions related to inclusion and exclusion criteria for the study.

## 2. Survey Completion Confirmation:

- 2.1 Upon completing the survey, participants will receive an automated email confirming their submission
- 2.2 The email will include a link to schedule a 30-minute virtual pre-screen interview via Google Meet on a HIPAA compliant version of Google Meet.

# 3. Pre-Screen Interview and Eligibility:

- 3.1 A licensed clinical social worker will conduct the pre-screen interview via Google Meet.
- 3.2 During the interview, the clinician will review the study procedures, timeline, and eligibility criteria with the participant.
- 3.3 Any questions or concerns the participant may have regarding the study will be addressed.
- 3.4 The clinician will assess the participant's eligibility based on the inclusion and exclusion criteria outlined in the study protocol.
- 3.5 If the potential participant does not meet the eligibility criteria, they will be informed during the phone call and given time to process their reaction. Specific details as to why they do not qualify will not be provided to prevent attempts to alter responses.
- 3.6 In cases where eligibility is unclear, the clinician will inform the potential participant that they will receive a follow-up email or phone call once their eligibility status is confirmed.
- 3.7 The clinician will then review with PI regarding eligibility. Once eligibility is confirmed, the clinician will set up a call to let the participant know the results. They will then go through the informed consent process.
- 3.8 If a participant does not meet criteria for the study and the PI has confirmed they do not qualify, the prescreen questionnaire will be permanently and securely deleted from the HIPAA compliant platform JotForm.
- 3.9 The clinician will read a script at the beginning of the pre-screen so that each potential participant is fully informed before beginning the process.
- \*See Appendix B for Prescreen Script

#### 4. Compliance and Review:

- 4.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 4.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 4.3 Research team will meet weekly to review study procedures, timeline, and compliance.

# iii. Title: Standard Operating Procedure for Participant Enrollment


Effective Date: [5.8.24] Review Date: [5.8.24]

**Objective:** To outline the process for participant enrollment for the Akashic Record Research Study in accordance with Institutional Review Board (IRB) guidelines, ensuring compliance with ethical standards and participant safety.

**Scope:** This procedure includes all those involved in the enrollment process; Co PI/Independent Evaluator and Research Coordinator

#### 1. Informed Consent Process:

- 1.1 If the participant meets eligibility criteria, the clinician will provide them with a copy of the informed consent form (ICF) and review it in detail.
- 1.2 Participants will have the option to sign the ICF electronically using Jotform during the pre-screen interview.
- 1.3 Alternatively, participants may choose to keep the ICF to review at their own pace and sign it electronically at a later time, but prior to any data collection activities. Research will not begin unless the client signs and returns the consent form.
- 1.4 The participant will be explained the protocol, time requirement, assessment scale types, session details, risk and benefits, staff roles and support, and all other components as outlined in the informed consent.
- 1.5 Clinician will use a checklist and script to present and review the informed consent in a consistent and ethical manner, with emphasis on voluntary participation.
- 1.6 Participants will be encouraged to reach out to the clinician with any additional questions or concerns regarding participation in the study.
- 1.7 During the ICF process, the clinician will read a script to participants before reading through the informed consent.
- \*See Appendix B for Prescreen and Informed Consent Script
- \*See Appendix C for Prescreen Checklist

#### 2. Scheduling Akashic Record Sessions

- 2.1 Once enrolled and the ICF has been signed, participants will receive guidance from the clinician on scheduling their Akashic Record sessions with the practitioner, Candice Rasa on Google Calendar through Google Workspace
- 2.2 The clinician will send participants a digital billing form via Google Workspace.
- 2.3 The clinician will then schedule both Akashic Record sessions with the client in Google Calendar The clinician will make sure the visits are scheduled within the protocol study timeline.
- 2.4 Participants will be reminded of the study schedule and the importance of staying within the timeframe. They will be reminded of the self-report scales and the timeline that they must be completed by.

#### 3. Enrollment and Unique Identification Number Assignment:

- 3.1 Upon signing the ICF and officially enrolling in the study, participants will be assigned a unique identification number (see SOP on Unique Identification Number for more information).
- 3.2 This unique identification number will serve as the primary identifier for the participant throughout the study.

## 4. Participant Communication

- 4.1 Clinician will send a follow up email to participant within 24 hours that includes session date confirmation, copy of signed informed consent, and contact information of study staff and IRB.
- 4.2 Research Coordinator will send email to participant within 7 to 10 days of first Akashic Session with links to initial clinical scales, Akashic prep form, and demographic form.

#### 5. Compliance and Review:

- 5.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 5.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 5.3 Research team will meet weekly to review study procedures, timeline. and compliance.

#### iv. Title: Standard Operating Procedure for Assigning Unique Identification Numbers


. \_

Effective Date: [5.8.24]

Review Date: [5.8.24]

**Objective:** To assign unique identification numbers to participants enrolled in the study, ensuring proper tracking and organization of participant data across various platforms while maintaining HIPAA compliance.

Scope: This procedure includes Co-PI/ Independent Evaluator

<sup>\*</sup>See Appendix D for Email Templates

## 1. Participant Enrollment:

1.1 Once a participant has signed the informed consent form and officially enrolled in the study, they will be eligible for assignment of a unique identification number.

#### 2. Unique Identification Number Assignment:

- 2.1 Assign a unique identification number to each participant, starting with "0001" and increasing numerically with each new participant enrolled Ex: "0002", "0003" etc.
- 2.1 Record the participant's name and assigned identification number in a spreadsheet on Jotform.
- 2.3 Utilize a HIPAA-compliant version of Jotform for the spreadsheet to ensure data security and compliance.

## 3. Integration with Google Workspace

- 3.1 Add the assigned unique identification number to the participant's profile in Google Workspace, along with their full legal name.
- 3.2 Ensure that all participant data in Google Workspace is updated to include the unique identification number for proper tracking and management.

## 4. Use of Unique Identification Number:

- 4.1 The assigned unique identification number will serve as the primary identifier for each participant throughout the study.
- 4.2 Utilize the unique identification number in all storage of recorded data, including recordings of Akashic sessions and interviews.
- 4.3 Ensure that the unique identification number is consistently used across all platforms and documentation related to the study.

#### 5. Compliance and Review:

- 5.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 5.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 5.3 Regularly review and update procedures to ensure compliance with HIPAA regulations and data security standards.
- 5.4 Maintain strict confidentiality of participant information and ensure secure storage of all data.

## v. Title: Standard Operating Procedure for Recording and Storage of Akashic Sessions


Effective Date: [5.8.24] Review Date: [5.8.24]

**Objective:** This Standard Operating Procedure (SOP) outlines the procedures for the recording and storage of data, subject to the Health Insurance Portability and Accountability Act (HIPAA) regulations.

**Scope:** This SOP applies to PI and Research Coordinator

#### **Responsibilities:**

- 1. Principal Investigator (PI):
  - 1.1 Ensures compliance with HIPAA regulations and IRB policies.
  - 1.2 Provides oversight of the recordings and storage process.

#### 2. Research Team:

- 2.1 Follow the procedures outlined in this SOP.
- 2.2 Report any concerns or incidents related to data security.

#### **Procedure:**

- 3. Informed Consent:
- 3.1 Obtain informed consent from all participants, clearly outlining the recording process, purpose, and potential risks.

## 4. Preparation:

- 4.1 Ensure all devices are password protected
- 4.2 Ensure all devices (phone, computer) are powered on and functioning properly.
- 4.2 Open Google Meet and verify HIPAA compliance.
- 4.3 Access Google Workspace's Drive and ensure proper permissions and compliance settings are in place.

## 5. Conducting the Session:

- 5.1 Begin the Akashic Record session with the participant.
- 5.1 Use the Google Meet platform for conducting the session, ensuring adherence to HIPAA guidelines and maintaining confidentiality.

#### 6. Post-Session Procedures:

- 6.1 Once the session is completed, stop the recording on the Google Meet.
- 6.1 Recordings will automatically transfer to a designated password protected cloud storage Google Workspace's Drive.
- 6.3 Verify that the recording is stored securely in compliance with HIPAA regulations.
- 6.4 Once per week, the Research Coordinator will make a second copy of all new recordings from the drive onto an encrypted jump drive for additional security.

#### 7. De-identification:

- 7.1 Remove any identifiable information from recordings before analysis.
- 7.2 Assign unique identifiers to participants for linkage with other study data.

## 8. Distribution of Recordings:

- 8.1 Access the recorded session in Google Workspace's Drive.
- 8.2 Prepare an email to the participant via Google Workspace.
- 8.3 Include a link to their specific recording in the email.
- 8.4 Ensure the link is accessible for 7 days to allow the participant to download the recording.
- 8.5 Send the email to the participant.

#### 9. Record Retention:

- 9.1 Maintain recordings of Akashic sessions for a period of 6 years on an encrypted jump drive.
- 9.2 Once the study is complete and all Akashic sessions have been conducted and stored on an encrypted jump drive, the recordings will be permanently deleted from google drive.
- 9.3 Regularly review and update storage protocols to ensure compliance with any changes in regulations or best practices.
- 9.4 After the retention period, securely delete recordings in accordance with data disposal procedures.

## 10. Reporting Incidents:

- 10.1 Report any unauthorized access, disclosure, or data breaches promptly to the IRB and relevant authorities.
- 10.2 Address the unauthorized access according to the incident response procedures and IRB regulations.

## 11. Training:

11.1 Provide training to all research team members on HIPAA regulations, data security, and the procedures outlined in this SOP.

#### 12. Document Control:

12.1 Maintain a record of all changes made to this SOP, including version updates.

#### 13. Data Collection:

- 13.1 Use encrypted and password-protected recording devices to capture the recording.
- 13.2 Minimize the collection of unnecessary personal information.
- 13.3 Ensure recording only captures data relevant to the research objectives.

#### 14. Data Storage:

- 14.1 Store recording on a secure, password-protected server or cloud storage system.
- 14.2 Use encryption protocols (e.g., AES-256) for data at rest.
- 14.3 Regularly backup recording to prevent loss and facilitate recovery.

#### 15. Access Controls:

- 15.1 Limit access to recordings data to authorized personnel only.
- 15.2 Assign unique user credentials for each team member and maintain an access log.

#### 16. De-identification:

- 16.1 Remove any identifiable information from recordings before analysis.
- 16.2 Assign unique identifiers to participants for linkage with other study data.

#### 17. Data Retention and Disposal:

- 17.1 Establish a clear data retention policy, specifying the duration recordings will be stored.
- 17.2 Develop procedures for secure data disposal when it is no longer needed for research.

#### 18. Reporting Incidents:

18.1 Report any unauthorized access, disclosure, or data breaches promptly to the IRB and relevant authorities.

#### 19. Training:

19.1 Provide training to all research team members on HIPAA regulations, data security, and the procedures outlined in this SOP.

## 20. Compliance and Review:

- 20.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 20.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 20.3 Research team will meet weekly to review study procedures, timeline. and compliance.

## vi. Title: Standard Operating Procedure for Participant Completion of Clinical Scales


Effective Date: [5.8.24] Review Date: [5.8.24]

**Objective**: This Standard Operating Procedure (SOP) outlines the procedures for participants to complete clinical scales, including the Depression Anxiety Stress Scales (DASS), the Warwick-Edinburgh Mental Well-being Scale (WEMWBS), and the Connor-Davidson Resilience Scale (CD-RISC 10).

**Scope**: This SOP applies to all participants involved in research studies requiring completion of clinical scales.

#### **Responsibilities:**

- 1. Study Coordinator:
- 1.1 Coordinate the distribution of clinical scales to participants.
- 1.2 Ensure participants receive clear instructions and adequate timeframes for completing the scales.
- 1.3 Monitor the completion status of scales and notify the research team upon completion.
- 2. Research Team:
- 2.1 Provide support to participants in completing the clinical scales, if needed.

2.2 Ensure timely review of completed scales and integrate data into the study database.

#### 3. Procedure:

- 3. Scale Distribution:
- 3.1 Study Coordinator will email participants a link to the appropriate scale along with the timeframe based off study timeline..
- 3.2 The email will specify the deadline by which participants must complete the scales.

## 4. Scale Completion:

- 4.1 Participants will click on the provided links in the email, which will direct them to the appropriate forms on JotForm.
- 4.2 Participants will fill out the self-report scales on JotForm, ensuring all required fields are completed before submitting.
- 4.3 Upon completion, participants will submit the forms electronically.

#### 5. Data Collection:

- 5.1 Study Coordinator will regularly monitor JotForm responses to track participant completion of scales.
- 5.2 Completed scales data will be securely stored and managed according to research protocol and regulatory requirements.

## 6. Notification of Completion:

- 6.1 Once participants complete the scales, the study coordinator will receive an automated email notification from JotForm.
- 6.2 The research team will review the completed scales and acknowledge receipt.

#### 7. Reporting Incidents:

7.1 Report any unauthorized access, disclosure, or data breaches promptly to the IRB and relevant authorities.

#### 8. Compliance and Review:

- 8.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 8.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 8.3 Research team will meet weekly to review study procedures, timeline. and compliance.

## vii. Title: Standard Operating Procedure for Scheduling, Recording, and Storing Virtual Interviews


Effective Date: [5.8.24] Review Date: [5.8.24] **Objective:** To conduct virtual interviews efficiently and securely using Google Calendar, Google Meet, and Google Drive while ensuring compliance with HIPAA regulations for the handling of Protected Health Information (PHI). Additionally, to ensure the secure collection of interview responses using JotForm.

**Scope:** This procedure involves Co-PI and Research Coordinator

**Interview Process:** The research team will conduct structured interviews with participants with the aim of completing between 30 to 50 interviews. The decision to stop interviewing will be made collectively by the research team. This decision will be based on identifying redundancies in participant responses, indicating saturation of data. Regular meetings will be held to assess the progress of interviews and determine if additional interviews are necessary.

#### 1. Schedule the Interview:

- 1.1 Access Google Calendar and create interview time slots for participants to sign up for.
- 1.2 Participants will be encouraged to select a time slot. Once they have selected one on Google Calendar, they will be emailed a link with the designated time and date.
- 1.3 Set the event's visibility to "Private" to ensure confidentiality.

#### 2. Conduct the Interview:

- 2.1 Join the scheduled Google Meet session at the designated time.
- 2.1 Verify that the correct participant is present and ready for the interview.
- 2.3 Ensure the participant is in a quiet and confidential space in which they can freely share personal information.
- 2.4 Review informed consent and interviewing procedures with the participant.
- 2.5 Conduct the interview while adhering to professional standards and maintaining confidentiality.

#### 3. Record the Interview:

- 3.1 Inform all participants that the interview is being recorded for documentation purposes.
- 3.2 Ensure that Google Meet settings allow only authorized users to join the meeting and that anonymous guests are not permitted.
- 3.3 Start recording the Google Meet session once a verbal confirmation has been given by the participant to begin recording (see semi-structured interview form for more details).

#### 4. Store the Recording:

- 4.1 After concluding the interview, stop the recording on Google Meet.
- 4.2 Access Google Drive and navigate to the appropriate folder for storing interview recordings.
- 4.3 Upload the recorded interview to Google Drive, ensuring it is stored securely.

- 4.4 Title the stored recording with participant's unique identifier number which is assigned after enrollment into the study
- 4.5 Configure access permissions on Google Drive to restrict access to authorized personnel only.
- 4.6 Once per week, the Research Coordinator will make a second copy of all new recordings onto an encrypted jump drive for additional security

## **5. Secure Collection of Interview Responses:**

- 5.1 After the interview, interview responses will be written down in a secure platform using JotForm, a password-protected website.
- 5.2 Any names or identifiable information will be removed from the interview transcriptions.
- 5.3 A paid subscription JotForm account, compliant with HIPAA regulations for the collection and storage of PHI, will be utilized.
- 5.4 Access to JotForm will be restricted to the research team, including the interviewer, who will have unique login credentials.
- 5.5 The practitioner conducting the interview will not have access to JotForm, ensuring additional security and privacy of collected interview responses.

## **6. Ensure HIPAA Compliance:**

- 6.1 Confirm that all necessary Business Associate Agreements (BAAs) with Google are signed and in place.
- 6.2 Ensure that PHI information is permitted under the HIPAA BAA.
- 6.3 Limit PHI exposure within the organization by setting calendar entries containing PHI to "Private" and restricting access to authorized personnel only.

#### 7. Retention and Access Control:

- 7.1 Once the study is complete and all interviews have been conducted, transcribed onto Dedoose and a backup is stored on an encrypted jump drive, the recordings will be permanently deleted from google drive.
- 7.2 Maintain interview recordings in an encrypted jump drive for the required retention period of 6 years.
- 7.3 Regularly review access controls and permissions on Google Drive to ensure compliance with HIPAA regulations.

#### 8. Reporting Incidents:

- 8.1 Report any unauthorized access, disclosure, or data breaches promptly to the IRB and relevant authorities.
- 8.2 Address the unauthorized access according to the incident response procedures and IRB regulations.

#### 9. Compliance and Review:

- 9.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 9.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 9.3 Research team will meet weekly to review study procedures, timeline. and compliance.

## viii. Title: Standard Operating Procedure for Qualitative Analysis of Structured Interviews


Effective Date: [5.8.24] Review Date: [5.8.24]

## **Objective:**

The purpose of this Standard Operating Procedure (SOP) is to ensure a systematic and thorough qualitative analysis of structured interviews conducted during research projects. The goal is to extract meaningful insights from participant responses through a rigorous analytical process.

**Scope:** This procedure involves Co-Pi and research staff

#### 1. Transcription:

- 1.1 Each interview will be transcribed verbatim onto JotForm or a similar platform for documentation purposes.
- 1.2 The transcriptions will be reviewed for accuracy and completeness before proceeding to analysis.

#### 2. Data Management:

- 2.1 Transcribed interviews will be imported into Dedoose, a secure, password protected qualitative data analysis software.
- 2.2 The research team will ensure that all transcriptions are securely stored and backed up to prevent data loss.

#### 3. Coding Process:

- 3.1 Two members of the research team will independently code the transcriptions using predefined codes or categories based on research objectives.
- 3.2 Coders will mark segments of text that correspond to specific themes, concepts, or categories identified in the interview responses.
- 3.3 Coding will be conducted systematically to ensure consistency and reliability in the analysis process.

#### 4. Inter-Coder Reliability:

- 4.1 After independently coding the interviews, the two coders will meet to compare and discuss their coding decisions.
- 4.2 Any discrepancies or differences in coding will be addressed through consensus-building discussions.
- 4.3 Consensus on coding decisions will be reached through open dialogue and agreement between coders

## 5. Theme Development:

- 5.1 Following the coding process, themes will be identified based on recurring patterns, topics, or concepts across the interviews.
- 5.2 Themes will be derived from the coded data and will reflect the main findings and insights from the interviews.
- 5.3 Each code will be categorized under relevant themes to facilitate data interpretation and analysis.

## 6. Documentation and Reporting:

- 6.1 All coding decisions, themes, and analytical insights will be documented systematically.
- 6.2 A comprehensive report will be prepared summarizing the key findings, themes, and implications of the qualitative analysis.
- 6.3 The report will be shared with relevant stakeholders and utilized to inform further research or decision-making processes.

## 7. Quality Assurance:

- 7.1 Regular quality checks will be conducted throughout the analysis process to ensure the integrity and validity of the data.
- 7.2 Documentation of the analysis process will be maintained to enable auditability and reproducibility of results.

#### 8. Compliance and Review:

- 8.1 The qualitative analysis process will adhere to all ethical guidelines and regulations governing research involving human participants.
- 8.2 Confidentiality and anonymity of participants will be maintained throughout the analysis process.
- 8.3 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 8.4 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 8.5 Research team will meet weekly to review study procedures, timeline. and compliance.

This SOP provides a structured framework for conducting qualitative analysis of structured interviews, ensuring consistency, reliability, and rigor in the interpretation of participant responses. By following these guidelines, the research team can derive meaningful insights to address research objectives and contribute to the body of knowledge in the relevant field.

# ix. Title: Standard Operating Procedure for Managing Conflict of Interest in a Study Measuring the Effectiveness of Akashic Record Sessions


Effective Date: [5.8.24] Review Date: [5.8.24]

**Objective:** Includes all those on the research team involved in ethics, procedure compliance and role and responsibilities of staff.

**Introduction:** This Standard Operating Procedure (SOP) outlines the protocol for managing conflicts of interest. To ensure the integrity and objectivity of the research, measures will be implemented to mitigate potential conflicts of interest.

## 1. Roles and Responsibilities:

- 1.1 Candice Rasa: Sponsor and interventionist.
- 1.2 Research Team: Responsible for data collection, analysis, and reporting.

#### 2. Data Access Restrictions:

- 2.1 Candice Rasa will not have access to any outcome related data to prevent potential bias or influence on the study outcomes until the study has completed.
- 2.2 Candice will not have access to JotForm, where the participant's self-report assessment scores are collected.
- 2.3 Candice will not have access to Dedoose, where semi-structured interview responses are stored.
- 2.4 The recordings of the interviews will be kept in a password protected folder on Google Workspace and Candice Rasa will not have permission to view them.

#### 3. Participant Communication:

- 3.1 Participants will be informed during the informed consent process that Candice Rasa, the sponsor and interventionist, will not have access to their self-report assessment scores.
- 3.2 This information will be communicated to participants to ensure transparency and prevent any potential bias or influence on their reporting behavior.
- 3.3 Participants will be encouraged to provide honest and accurate responses during the assessment process, knowing that their scores will not be accessible to Candice Rasa.

#### 4. Access Permissions:

4.1 Candice Rasa will only have access to certain folders in Google Workspace which is a platform containing participant names and unique identification numbers.

4.2 Access will be limited to participant identification information necessary for scheduling and session management.

## 5. Data Handling Procedures:

- 5.1 The research team will ensure strict adherence to data access restrictions and handling protocols.
- 5.2 All data will be secured with appropriate access controls and encryption measures.
- 5.3 Research Coordinator will be responsible for monitoring access permissions
- 5.4 Co-investigator will be responsible for assigning UIN for research participants

## 6. Confidentiality Measures:

- 6.1 Confidentiality agreements will be signed by all research team members, including Candice Rasa, to uphold participant privacy and data confidentiality.
- 6.2 Participant identifiers will be anonymized in all analysis and reporting to maintain confidentiality.

## 7. Training and Awareness:

- 7.1 All research team members will receive training on conflict of interest policies and procedures.
- 7.2 Ongoing awareness efforts will be implemented to promote transparency and ethical conduct throughout the study.

## 8. Reporting and Documentation:

- 8.1Any instances of potential conflicts of interest or breaches of protocol will be promptly reported to the oversight committee.
- 8.2 Comprehensive documentation of data access, handling, and decision-making processes will be maintained for audit and review purposes.

#### 9. Transparency and Disclosure:

- 9.1 Any potential conflicts of interest involving Candice Rasa will be disclosed in study publications and reports.
- 9.2 Transparency will be maintained in all aspects of the study to ensure the integrity and credibility of the research findings.

#### 10. Compliance and Review:

- 10.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 10.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.

10.3 Research team will meet weekly to review study procedures, timeline. and compliance.

## x. Title: Standard Operating Procedure for Participant Withdrawal from Study


Effective Date: [5.8.24] Review Date: [5.24.24]

**Objective:** To establish a protocol for handling participant withdrawal from the study, ensuring the integrity of collected data and maintaining participant confidentiality while allowing for optional continued follow-up.

**Scope:** This procedure applies to all studies involving subjects undergoing Akashic Record sessions with Candice Rasa LCSW, with provisions for participant withdrawal and optional continued follow-up for mental health outcome assessments.

#### 1. Data Retention:

1.1 Data collected on the participant up to the point of withdrawal must remain part of the study database and cannot be removed.

#### 2. Discussion on Continued Follow-up:

- 2.1 If the participant withdraws from the interventional portion of the study, they will not be sent or asked to complete any further self-report assessments and their participation in the trial will end
- 2.2 Investigators are responsible for initiating and facilitating discussions with withdrawing subjects to discuss confidentiality of their data and address any concerns.

#### 3. Eligibility for Reentry:

- 3.1 Participants who have previously withdrawn from the study may express interest in reentering at a later time.
- 3.2 However, participants who have completed one or both of the Akashic Record sessions are ineligible for reentry due to issues with the study timeline.

#### 4. Review of Study Data and Public Records:

4.1 The investigator may review study data related to the participant collected prior to the withdrawal.

## 5. Compliance and Review:

- 5.1 This SOP will be reviewed and approved by the IRB to ensure compliance with ethical standards and participant safety.
- 5.2 Regular audits and assessments will be conducted to ensure ongoing adherence to the SOP and IRB guidelines.
- 5.3 Research team will meet weekly to review study procedures, timeline. and compliance.

#### APPENDIX B

## **Scripts**

## **Prescreen Script:**

Hello and thank you for considering joining our study. Before we begin, I'd like to explain the purpose of this interview. The goal of this interview is to see if you're a good fit for the study.

Doing this interview is voluntary. You have the right to stop the interview at any time.

Your privacy is important to us. Any information you share during this interview will be kept private. Your responses will only be used to see if you meet the criteria. If you choose not to participate in the study or if you can't participate, your information will be deleted.

If at any point during the interview you feel uncomfortable or wish to stop, please let me know. We will end the interview right away.

With that said, are you ready to begin the interview?

#### **Informed Consent Script**

"Thank you for your interest in participating in our research study. I want to ensure that you have all the information you need to make an informed decision about joining this study. We will be going over the informed consent form together, which outlines the purpose, procedures, risks, and benefits of the study. I'll be reading through the entire informed consent document with you. Please feel free to stop me at any time if you have any questions or need clarification. It's important for you to know that your participation in this study is entirely voluntary. If at any point you decide you no longer wish to participate, that's okay, and there won't be any consequences. You may also keep the informed consent and review it at home, privately. Take as much time as you need to decide if you wish to participate. You are not required to sign the informed consent today."

## **Akashic Prep Discussion Script:**

Thanks for joining our research on Akashic Records! Today, I'll explain what we'll be doing and what you can expect. The Akashic Records are like a special library in the universe that holds all sorts of information about your soul, like your past lives, the patterns you follow, and even things from your ancestors. Because your soul isn't physical and doesn't disappear, the memories inside it can be accessed and read. Anyone can learn to read these records. When we start, I'll be like a translator. You'll ask questions, and I'll get pictures, words, feelings, and thoughts that I'll share with you. It works best if you focus on how things feel rather than trying to figure everything out in your head. For example, if I tell you something, try to feel it in your heart and body and think about how it connects to your life. It's okay to feel emotional during our session. We'll begin with an introduction that will last about 5 to 10 minutes. Please wait until it's finished to ask questions, so you get all the information. If something makes you feel emotional, make a note of it, because you might want to ask about it later. You can write things down if you want, but just listening and feeling is the best way to understand. After the intro, we'll talk about what came up for you. Then, we can focus on whatever you're interested in. I suggest asking about things that trigger feelings of anxiety, stress, or depression or things that keep happening in your life. You can also ask about people close to you, but we'll focus on what you're meant to learn from them, not just gossip about their lives. I'm here to help you, so feel free to ask anything you need. Do *you have any questions?* 

## **Akashic Session Completion Script:**

I hope you found today's information helpful. I suggest listening to the recording of our session at least once before our next meeting. Sometimes we understand things better the second time we hear them. It's a good idea to take some time to rest and think about what we talked about. You can also talk to someone you trust to help you understand it better. If I gave you any suggestions or resources, you can start with the ones that sound most interesting to you. You don't have to do everything right away. Listen to your heart and start with what feels right. It might be helpful to keep a little journal of any thoughts or questions you have so you can ask them in our next session. Do you have any questions about that?

Remember to fill out the three self-assessment scales for our research study. We'll email you the links for them soon. Also, just so you know, I won't be able to see your answers to the scales during the study. If you have any questions about the scales or anything else, you can ask Betsy, our research coordinator, or Sarah, the independent evaluator.

#### **Semi-Structured Interview Script and Questions:**

**Thank you and purpose:** Thank you for doing this study. As you know, this study is about how two Akashic Record sessions impact mental health. We want to know how a person's connection to self and connection to others is impacted by a session. We are also interested to see how their view of anxiety, stress and depression changes after having two sessions. Our goal is to learn more about what parts of Akashic Record sessions people may find helpful for them.

Confidentiality: We will summarize the answers of all the participants in this study. Your individual answers will not be shared with anyone. It is in your rights to recall your consent at any time. I want to be sure that you are comfortable with this process, and that you understand you may stop me at any time during the interview. All the information you share will not be shared with anyone. To keep things confidential, we will remove all names that may come up during the interview.

**Recording:** You gave your consent to be recorded. If you wish to explain something and not be recorded, please let me know at that time and I will stop the recording.

INTERVIEWER: [Start recording]

I will ask you questions about your experience with the Akashic Record sessions you had with Candice Rasa. I will start by asking questions about why you joined this study. I will then ask about what you found helpful and what new ideas you got from it. I will then ask you questions about what part of the sessions you found to be difficult or any challenges you have found integrating what you learned into your daily life.

We want to know your honest opinions and experiences. In answering the questions, we would like you to provide as many details as you can to help us understand your experiences. Please remember that there is no right or wrong answer to any of these questions, and your individual answers will not be shared with anyone.

#### **Participation**

1. What motivated you to seek help through the Akashic Record sessions? [Areas for probing: What did you want to improve or work on? What were you hoping or expecting to get out of these Sessions?]

#### The Akasha

2. Did you know about the Akasha before joining in this study? [Areas for probing: Can you share more about how your understanding of the Akasha has changed over the course of the 2 sessions provided?]

#### **Benefits**

- 3. Thinking back on your experiences, what parts of the sessions did you find most helpful?
- 4. Can you share about your view of your challenges or problems compared to before you started this study? [Areas for probing: Can you share any specific insights you gained during the sessions that helped you in working on your challenges?]

## Integration

- 5. How has the process been for you since your second session? How has it been integrating the new insights that you got from the sessions into your daily life?
- 6. Can you share whether you used the interventions or practices that were suggested to you during your session? Why or why not?

## Challenges

7. Were there any other difficulties you faced during or after the sessions? If so, can you share some details about those experiences?

# APPENDIX C Staff Checklists

#### **Phase 1: Application and Approval Process**

Participant seeks information about research study

- Participant reads information about research study via world of mouth, on landing page, or social media post
- Participant clicks link to prescreen application housed on Jotform

Participant completes prescreen steps

- Participant completes prescreen application on Jotform
- Schedules self for prescreen interview with Sarah Coleman by clicking hyperlink to Google Meet

Sarah Coleman completes prescreen interview

| Conducts prescreen | interview with | h participant | via Goog | gle Meet |
|----------------------|----------------|---------------|----------|-----------|
| Determines eligibili | ty + consults | with Candice | Rasa as | necessary |

| ☐ Reviews study timeline with participant |
|---|
| ☐ Emails ICF to participant to review |
| ☐ Reviews and signs ICF with participant |
| ☐ Sets Akashic Appointments for participant in Google Meet |
| ☐ Sends participant billing form |
| ☐ Explains two options (payment plan) and explains that the session must be paid for before the first session |
| ☐ Sends confirmation email with session dates + timeline + ICF to participant |
| ☐ Assigns unique number to participant in Jotform |
| ☐ Remind participant of next step |
| ☐ Add steps completed into Monday |
| Betsy Koczab sends study documents to participant |
| ☐ Demographic form (Jotform) |
| ☐ 1st set of scales (Jotform) |
| Phase 2: Self Assessments and Akashic Session |
| Candice Rasa completes initial 90 min Akashic Session |
| ☐ Completes initial Akashic Assessment |
| ☐ Reminds participant of upcoming scales |
| ☐ Remind participant of next step |
| Betsy Koczab sends follow-up documents to participant |
| ☐ Emails participant session recording link |
| ☐ Backs up session recordings to jump drive |
| ☐ Sends links to 2nd set of scales |
| Candice Rasa completes follow-up 50 min Akashic Session |
| ☐ Completes follow-up Akashic session |
| ☐ Reminds participant of upcoming scales |
| ☐ Schedules participant for semi-structured interview with Sarah Coleman in Google Meet |
| ☐ Remind participant of next step |
| Betsy Koczab sends follow-up documents to participants |
| ☐ Emails participant session recording link |

| ☐ Backup session recordings to jump drive |
|---|
| ☐ Sends links to 3rd set of scales |
| ☐ Send link to satisfaction survey |
| ☐ Inputs 60 day follow-up date in Monday.com (set as 60 days from 2nd Akashic Session) |
| Phase 3: Final Assessments and Semi-structured Interview |
| Sarah Coleman completes semi-structured interview |
| ☐ Conducts structured interview in Google Meet |
| ☐ Transcribes interview in Jotform |
| ☐ Remind participant of last set of scales in 2 months |
| Betsy Koczab completes participant from study |
| ☐ Backs up semi structured interview to jump drive |
| ☐ Sends thank you email to participant that includes ongoing mental health referrals |
| ☐ Betsy sends email to participant to complete 4th set of scales at 60 day follow-up |
| APPENDIX D Templates |
| Recruitment Templates |
| Landing Page + Email Marketing |
| Subject: A Call For People To Join |
| Hello First name / friend |
| Good news! We're inviting people to join our Akashic Research study. |
| Here, you can learn about the research and start to apply. |
| Research Title: Exploring How Akashic Records Affect Mental Health |
| <b>Research Goal:</b> We want to see if Akashic Records can help people who feel stressed, anxious or depressed. |

**Our Question:** Can Akashic Records make people feel less stressed, sad, or anxious, and more resilient and connected?

What are the Akashic Records: Akashic Records are like a big library in space where all knowledge is kept. People who can tap into this library use special senses to understand and share the information. During sessions, they might talk about past lives, feelings, family history, and other personal stuff. They also offer advice and help tailed to the client's needs.

**Akashic Sessions:** Candice Rasa, LCSW, will lead the sessions. They will last about 50-90 minutes and you can schedule a session at a time that works for both you and Candice. You can decide what is talked about by asking questions about your life.

**Study Plan**: You'll have two Akashic Sessions: one session that is 90 minutes and one shorter follow-up session that is 50 minutes.. You'll also answer some questions on a form about your experience. At the end, you'll have an interview with Sarah Coleman, LCSW.

**Study Time:** The study will take about 3 months to complete.

Where: All sessions will be held online through a website called Simple Practice.

**Who Can Join:** You can join if you're 18 or older, have felt stressed, sad, or anxious in the past year, haven't had an Akashic Session with Candice Rasa LCSW before, and don't have problems with drugs, thoughts of hurting yourself, or serious mental health issues.

**Next Steps:** To join, please click the link below to fill out the application.

[link to Jotform prescreen]

This research is sponsored by Rasa Healing, Inc. Candice Rasa, LCSW, will lead the sessions, and Sarah Coleman, LCSW, will conduct the interviews.

#### **Contact Information:**

For questions or concerns regarding the study, you may contact Sarah Coleman at va.research@rasahealingservices.com or Candice Rasa at candice@rasahealingservices.com

An institutional review board (IRB) is an independent committee established to help protect the rights of research subjects. If you have any questions about your rights as a research subject, contact (Monday through Friday 9-5 EST/EDT):

By mail: Pearl IRB 29 East McCarty Street Suite 100 Indianapolis, IN 46225

https://www.pearlirb.com/

or call: 317-899-9341 (main) or fax: 317-602-6554 (fax)

or by email: <a href="mailto:support@pearlirb.com">support@pearlirb.com</a>

Please reference the IRB study number when contacting the IRB.

## **Social Media Posts**

Post #1

We're now (still) looking for volunteers for our Akashic Research study!

We want to see how Akashic Record sessions affect people who feel anxious, sad, or stressed.

You might be able to join if you're 18 or older, felt sad, anxious, or stressed in the past year, haven't had an Akashic Session with Candice Rasa LCSW before, and don't have problems with drugs, or thoughts of hurting yourself.

First, you'll read about the study and fill out a short form. You'll find out why we're doing this, what the study involves, how long it takes, and what Akashic sessions are like. To find out more and sign up, click the link in my bio.

We're really excited about this project! Please tell anyone who might want to join.

#### Post #2

If you're new to the Akasha and want to understand it better before joining our study, here's what it's all about:

The Akashic Record is like a big library in the sky where all information and knowledge is kept. People who can tap into this library are trained to sense and understand the information using special psychic abilities like seeing things in their mind (clairvoyance), hearing things in their head (clairaudience), just knowing things (claircognizance), and feeling things (clairsentience). They get information from this library and share it with others. During Akashic sessions, they might talk about past lives, emotional patterns, family history, and other personal stuff. They also offer advice and resources to help.

In our study, Candice Rasa, LCSW, will use her skills to tap into the Akashic Record for you. Each session will be about 50-90 minutes long and we'll find a time that works for both of us. You can decide what topics we talk about by asking questions about your life.

If you're interested in joining our study, the first step is to read more about it and fill out a short form. You'll learn why we're doing this, how the study works, what we expect, and what happens during Akashic sessions. Just click the link in my profile to learn more and sign up.

We're really excited to get started, and please tell others who might want to join too!

#### **Post #3**

We're doing this research because we want to understand how Akashic Records affect people's mental health. Here's what we're looking at:

Research Title: Studying How Akashic Records Sessions Affect Mental Health

**Research Goal:** We want to see how Akashic Records help people who feel stressed, sad, or anxious

**Our Question:** Can Akashic Records sessions make people feel less stressed, sad, or anxious, and more resilient and connected?

If you want to join our study, first, you need to read about it and fill out a short form. You'll learn why we're doing this, how it works, what we expect, and what happens during Akashic sessions. Just click the link in my profile to learn more and sign up.

We're really excited to get started, and please tell others who might want to join too!

## **Email Sequence Templates**

## Welcome Email: (sent by Co-PI Sarah Coleman)

Subject: You are enrolled: Akashic Research Study

Hi there (name)

Thank you for being part of our research. Your Akashic Sessions are scheduled for (date) and follow-up on (date). Please find the timeline for the study to help you stay on track attached. You will get an email from our Research Coordinator Betsy within 7 days of your Session. She will let you know when to complete your first self-report scale. These are time sensitive so please keep this in mind. They must be completed before your first session. Here are a couple of important points:

Please only use the links from our emails as we send them. Do not use links from old emails. Each self-report is connected to a specific report in the research timeline.

If you have a question about scheduling or scale completion, please reach out to our Research Coordinator, Betsy Koczab va.rasahealing@gmail.com. If you have a question about the Akashic Sessions, please contact Candice Rasa, LCSW at candice@rasahealingservices.com (name/ contact info)

## Akashic Research First Set of Scales: (sent by Betsy Koczab, Research Coordinator)

Subject: Subject: 1st Set of Scales READY: Akashic Research

Hi there (participant name)

You are now eligible to complete your 1st set of assessment scales.

These scales are necessary for you to begin your participation in Akashic Research. These forms are required *prior* to your Akashic Session with Candice.

Again, you can find them directly below:

- DASS scale, after 1st Akashic Session
- WATTS scale, after 1st Akashic Session
- CD-RISC 10 scale, after 1st Akashic Session
- Demographic form (one time only form)

You can access the prep form for your Akashic Session HERE. It is also attached. Please review it prior to your first Akashic Session.

Let me know if you have any questions about the process. I am here to support you and ensure successful engagement in the research.

(name/contact info)

#### Akashic Research Second Set of Scales: (sent by Betsy Koczab, Research Coordinator)

Subject: 2nd Set of Scales READY: Akashic Research

Hi there (participant name)

The recording from your initial Akashic Assessment can be found HERE [insert link] You are now eligible to complete the 2nd set of assessment scales entitled "After 1st Akashic Session"

You can found them below:

- DASS scale
- WATTS scale
- CD-RISC 10 scale

As a reminder, please use the above link for the 2nd set of assessment scales, versus prior emails, as these links are directly tied to #2 scales.

Let me know if you have any questions about the process. I am here to support you and ensure successful engagement in the research.

(name/contact info)

## Akashic Research Third Set of Scales: (sent by Betsy Koczab, Research Coordinator)

Subject: 3rd Set of Scales READY: Akashic Research

Hi there (participant name)

The recording from your follow-up Akashic Session can be found HERE [insert link]

You are now eligible to complete the 3rd set of assessment scales entitled "After 2nd Akashic Session"

You can found them below:

- DASS scale After 2nd Akashic Session
- WATTS scale After 2nd Akashic Session
- CD-RISC 10 scale After 2nd Akashic Session
- Satisfaction Survey (This is a one time survey, please complete it along with others)

As a reminder, please use the above link for the 3rd set of assessment scales, versus prior emails, as these links are directly tied to #3 scales.

Let me know if you have any questions about the process. I am here to support you and ensure successful engagement in the research.

(name/contact info)

## Akashic Research 60 Day follow-up:(sent by Betsy Koczab, Research Coordinator)

Subject: 60 Day Follow-up: Akashic Research

Hi there (participant name)

Thank you for participating in our Akashic Research study. There is one final set of scales to complete.

You are now eligible to complete the 4th set of assessment scales entitled "60 Day Follow-up" You can found them below:

- DASS scale
- WATTS scale
- CD-RISC 10 scale

As a reminder, please use the above link for the 4th set of assessment scales, versus prior emails, as these links are directly tied to #4 scales for the 60 day follow-up.

Let me know if you have any questions about the process. I am here to support you and ensure successful engagement in the research.

(name/contact info)

#### Completion of Study email: (sent by Betsy Koczab, Research Coordinator)

Subject: Thank You for Completing the Akashic Records Study

Dear [Participant's Name],

We want to take a moment to thank you for being a part of the Akashic Records study. Your involvement is important and will help us learn more about Akashic Record Sessions.

Now that the study is finished, we want to offer you more support. Attached to this email, you'll find a referral sheet. This sheet has extra resources and people who can help you based on your interests and needs.

If you want to keep working with Candice, you can visit her website here:

[Insert Candice's Contact Information]

If you're looking for individual therapy, you can also work with Sarah. You can reach out to her directly at:

[Insert Sarah's Email Address]

If you need services for mental health and personal growth, please see our attached extended referral list.

Your commitment to growing and exploring is really wonderful Thank you once again for your important contribution to our study.

## **Akashic Prep Template**

## **Preparing for your Akashic Session**

#### What to expect:

- The Akashic Records are a channeled practice, where I translate information from the Akashic Record and share it with you.
- During an Akashic Session, you ask questions about your life and I channel/translate spiritual information from the Akashic field for you.

## **Asking Questions:**

- You have the right to ask anything you want. However, questions supporting your highest and best healing are ideal. Please take the time to write questions in advance and bring them to the session. This helps to set the intention, tone and topics of your session
- It is best to ask one question at a time, rather than two questions in one sentence, this way you get clear and precise answers. You can always ask follow up questions in the moment on any answers you receive that you want more clarity on.
- List questions in order of importance so we ensure that all of your pressing questions are covered in the time slot.
- Please note that questions about other people's motives or intentions are outside of the boundaries and scope of the Akasha.

## Sample Questions-Feel free to add/delete or bring your own:

- What gifts or talents do I have from a past life that I am not currently utilizing in this life?
- What is my biggest block right now?
- What strength or asset do I have that is helping me with this block?
- What healthy or unhealthy patterns am I experiencing now?
- How can I heal or shift that pattern/block right now?
- What am I learning from my current relationship with (name of person)?
- Why am I so (feeling or fear you may have)?
- Can you show me a past life or pattern where my fear of comes from?
- How can I heal or shift my karmic relationship with (name of person)?
- I have been coping with (name of pattern here). Where does this pattern come from?
- I have been coping with (unexplained or persistent physical ailment or pain or emotional condition). Can you show me a past life where this stems from?
- What's the most important thing for me to know right?

## **Mental Health Referral Template**

## Mental Health Referral Sheet for Spiritual and Emotional Support

#### Find a Therapist' Online Directories

- Psychology Today: <a href="https://www.psychologytoday.com/us/therapists">https://www.psychologytoday.com/us/therapists</a>
- GoodTherapy.org: <a href="http://www.goodtherapy.org/find-therapist.html">http://www.goodtherapy.org/find-therapist.html</a>
- American Association for Marriage and Family Therapy: https://aamft.org/Directories/Find a Therapist.asp

#### Free therapy and support services:

- Therapy Aid Coalition: https://psychcentral.com/reviews/online-therapist-for-free#therapy-aid-coalition
- Bliss: <a href="https://psychcentral.com/reviews/online-therapist-for-free#bliss">https://psychcentral.com/reviews/online-therapist-for-free#bliss</a>
- DRK Beauty Healing: For nonbinary and people of color: https://psychcentral.com/reviews/online-therapist-for-free#drk-beauty-healing

#### Hotlines

- 988 Mental Health Emergency Hotline: Calling 988 will connect you to a crisis counselor regardless of where you are in the United States.
- National Alliance on Mental Illness (NAMI) HelpLine: 1-800-950-NAMI, or text "HELPLINE" to 62640. Both services available between 10 a.m. and 10 p.m. ET, Monday–Friday
- U.S. Department of Health and Human Services Substance Abuse Treatment referral hotline 1-800-662-HELP (4357)
- National Domestic Violence Hotline: 1-800-799-7233
- National Suicide Prevention Lifeline: 1-800-273-TALK (8255); www.suicidepreventionlifeline.org. Or, just dial 988
- Suicide Prevention, Awareness, and Support: www.suicide.org
- Self-Harm Hotline: 1-800-DONT CUT (1-800-366-8288)
- Family Violence Helpline: 1-800-996-6228
- Planned Parenthood Hotline: 1-800-230-PLAN (7526)
- National Council on Alcoholism & Drug Dependency: 1-800-622-2255
- LGBTO Hotline: 1-888-843-4564
- National Maternal Mental Health Hotline: 1-833-TLC-MAMA (1-833-852-6262)
- The Trevor Project: 1-866-488-7386 or text "START" to 678678. Standard text messaging rates apply. Available 24/7/365. (Provides crisis intervention and suicide prevention services to lesbian, gay, bisexual, transgender, queer & questioning—LGBTQ—young people under 25.)
- The SAGE LGBT Elder Hotline connects LGBT older people and caretakers with friendly responders. 1-877-360-LGBT (5428)
- The Trans Lifeline is staffed by transgender people for transgender people: 1-877-565-8860 (United States) 1-877-330-6366 (Canada)
- Rape Abuse and Incest National Network (RAINN) is the nation's largest organization fighting sexual violence: (800) 656-HOPE / (800) 810-7440 (TTY)
- Veterans Crisis Line: https://www.veteranscrisisline.net
- International Suicide Prevention Directory: findahelpline.com
- The StrongHearts Native Helpline is a confidential and anonymous culturally appropriate domestic violence and dating violence helpline for Native Americans, available every day from 7 a.m. to 10 p.m. CT. Call 1-844-762-8483.

## **Text and App Resources**

- Psychological First Aid: <a href="https://www.nctsn.org/resources/pfa-mobile">https://www.nctsn.org/resources/pfa-mobile</a>
- Crisis Text Line: Text REASON to 741741 (free, confidential and 24/7). In English and Spanish
- Meditation apps: Insight Timer, Calm, Headspace, Aura, 10 Percent Happier, Smiling Mind, Simple Habit, Oak, Unplug, Omvana